
## The GlaxoSmithKline group of companies

OTX116505

| Division | Worldwide Develop | ment |
|------------------|---------------------|----------------|
| Information Type | Reporting and Analy | sis Plan (RAP) |

| Title | ; | Reporting and Analysis Plan for Study OTX116505: A Single Blind, Randomised, Placebo Controlled, Repeat Dose, Dose Escalating Study Investigating Safety, Tolerability Pharmacokinetics, Pharmacodynamics and the Beta Cell Preserving Effect of Otelixizumab in New-Onset, Autoimmune Type 1 Diabetes Mellitus Patients. |
|---|---|---|
| Compound Number | * | GSK2136525 |
| Effective Date | 1 | 20/NOV/2018 |

# **Description:**

The purpose of this reporting and analysis plan (RAP) is to describe:

- The planned final analyses and output to be included in the Clinical Study Report for Protocol 2011N129686\_09
- Describe the safety, tolerability, pharmacodynamic, pharmacokinetic and efficacy analyses required for the study which will be provided to the study team members to convey the content of the reporting efforts, specifically Statistical Analysis Complete (SAC) end of study deliverable

# The GlaxoSmithKline group of companies

# RAP Author(s):

| Author | Date |
|---|---|
| Senior Biostatistician (Early Phase Biostatistics and Programming) | See PMED electronic signature at end |
| Statistics Leader (Clinical Statistics, Biostatistics) | 19-Nov-2018 |
| Job Title (Clinical Programming, Biostatistics) | 19-Nov-2018 |

# The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Investigation Lead (Immuno-<br>Inflammation Experimental Medicine Unit) | 14-Nov-2018 | Email |
| Biology Lead (Immuno-Inflammation<br>Experimental Medicine Unit) | 15-Nov-2018 | Email |
| Pharmacology Lead (Immuno-Inflammation,<br>Clinical Pharmacology Modelling & Simulation) | 15-Nov-2018 | Email |
| Data Quality Lead (Immuno-Inflammation,<br>Global Clinical and Data Operations) | 15-Nov-2018 | Email |
| Safety Lead (Immuno-Inflammation, Global Clinical Safety & Pharmacovigilence) | 19-Nov-2018 | Email |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Statistics Director (Clinical Statistics, Biostatistics) | 19-Nov-2018 | Email |
| Programming Manager (Clinical Programming, Biostatistics) | 19-Nov-2018 | Email |

Copyright, 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | INTRODUCTION | 7 |
| | 1.1. RAP Amendments | |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 11 |
| | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | 11 |
| | 2.2. Study Objective(s) and Endpoint(s) | 11 |
| | 2.3. Study Design | 14 |
| | 2.4. Statistical Hypotheses | 15 |
| 3. | PLANNED ANALYSES | 15 |
| | 3.1. Interim Analyses | |
| | 3.2. Final Analyses | |
| 4. | ANALYSIS POPULATIONS | 16 |
| | 4.1. Protocol Deviations | 18 |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONVENTIONS | 19 |
| | 5.1. Study Treatment & Sub-group Display Descriptors | 19 |
| | 5.2. Baseline Definitions | 19 |
| | 5.3. Other Considerations for Data Analyses and Data Handling Conventions | 20 |
| 6. | STUDY POPULATION ANALYSES | 21 |
| | 6.1. Overview of Planned Analyses | 21 |
| | 6.2. Exposure | 21 |
| | 6.3. Concomitant Medication and Insulin Usage | 21 |
| 7. | | 21 |
| | 7.1. Adverse Events Analyses | 21 |
| | 7.2. Adverse Events Related to CRS and EBV Reactivation | 22 |
| | 7.3. EBV Serology and Viral Load | 22 |
| | 7.4. Cardiovascular Events | 22 |
| | 7.5. Clinical Laboratory Analyses | 22 |
| | 7.6. Other Safety Analyses | 22 |
| 8. | PHARMACOKINETIC ANALYSES | 22 |
| | 8.1.1. Drug Concentration Measures | |
| | 8.2. Derived Serum Pharmacokinetic Parameters | 23 |
| 9. | EFFICACY ANALYSES | 24 |
| | 9.1. Overview of Planned Efficacy Analyses | 24 |
| | 9.1.1. Endpoints / Variables | 24 |
| | 9.1.2. Summary Measure | 24 |
| | 9.1.3. Population of Interest. | 24 |
| | 9.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | 9.1.5. Statistical Analyses / Methods | 25 |
| | 9.1.5.1. Statistical Methodology Specification - MMRM | 26 |

9.2. Overview of Planned Pharmacodynamic Analyses ......27

| | | 9.2.1. | Endpoints / Variables | 27 |
|---|---|---|---|---|
| | | 9.2.2. | Summary Measure | 28 |
| | | 9.2.3. | Population of Interest | 28 |
| | | 9.2.4. | Strategy for Intercurrent (Post-Randomization) Events | 28 |
| | | 9.2.5. | Statistical Analyses / Methods | 28 |
| | 9.3. | Pharmad | cokinetic / Pharmacodynamic Analyses | 28 |
| | 9.4. | Overviev | v of Planned Exploratory Analyses | 28 |
| | | 9.4.1. | Endpoints / Variables | 28 |
| | | 9.4.2. | Summary Measure | 28 |
| | | 9.4.3. | Population of Interest | 29 |
| | | 9.4.4. | Strategy for Intercurrent (Post-Randomization) Events | 29 |
| | | 9.4.5. | Statistical Analyses / Methods | 29 |
| | | 0.1.0. | Otationida / Trially 000 / Motrodo | |
| 10. | REFE | RENCES | | 30 |
| 11. | APPE | NDICES | | 31 |
| | 11.1. | | x 1: Schedule of Activities | |
| | | 11.1.1. | Protocol Defined Time & Events | |
| | | 11.1.2. | | |
| | | 11.1.3. | | 33 |
| | | 11.1.4. | Dosing and Follow-Up Detail for Vitals, ECG and PK & PD Monitoring over the | |
| | | I la la Ta | Infusion Period (Cohorts 1-4) | 36 |
| | 11.2. | Annendi | x 2: Assessment Windows | 38 |
| | 11.4. | 11.2.1. | Definitions of Assessment Windows for Analyses | 39 |
| | 11.3. | | v 3: Ctudy Dhacas | 39 |
| | 11.3. | 11.3.1. | x 3: Study Phases | |
| | | 11.0.1. | Study Phases | 30 |
| | 11.4. | Annondi | x 4: Data Display Standards & Handling Conventions | 38 |
| | 11.4. | 11.4.1. | Derivations and Handling of Missing Baseline Data | 40 |
| | | 11.4.2. | | 40 |
| | 44.5 | 11.4.3. | Reporting Standards | 41 |
| | 11.5. | | x 5: Derived and Transformed Data | |
| | | 11.5.1. | | |
| | | 11.5.2. | Study Population | 42 |
| | | 11.5.3. | Safety | |
| | | 11.5.4. | Efficacy | 47 |
| | A1111111111111111111111111111111111111 | 11.5.5. | Pharmacodynamics | |
| | 11.6. | | x 6: Premature Withdrawals & Handling of Missing Data | |
| | | 11.6.1. | | 52 |
| | | 11.6.2. | Handling of Missing Data | 53 |
| | | 11.6.3. | Handling of Partial Dates | 53 |
| | 11.7. | Appendi | x 7: Values of Potential Clinical Importance | 54 |
| | | 11.7.1. | Laboratory Values. | 54 |
| | | 11.7.2. | ECG | 55 |
| | | 11.7.3. | Vital Signs | 55 |
| | 11.8. | Appendi | x 8: Biomarker Analyses | 56 |
| | | 11.8.1. | Handling of duplicate data due to reruns | 56 |
| | | 11.8.2. | Frequency and phenotype of lymphocyte subsets by flow | |
| | | | cytometry | 56 |
| | | 11.8.3. | Percentage of CD3 cells, FoxP3 regulatory cells and TH17 | 50 <del>-2.00</del> |
| | | | cells by epigenetic quantification | 58 |

## CONFIDENTIAL

# OTX116505

| | 11.8.4. | Frequency and phenotype of HLA-A2-resticted antigen- | |
|---|---|---|---|
| | | specific CD8+ T cells by multimer analysis | 59 |
| | 11.8.5. | Frequency of interferon-gamma- secreting antigen- | |
| | | reactive cells by ELISPOT | 62 |
| | 11.8.6. | Quantification of serum cytokines and soluble cytokine | |
| | | receptors. | 63 |
| | 11.8.7. | TCR deep sequencing | 64 |
| | 11.8.8. | Suppressive activity of regulatory cells | 65 |
| | 11.8.9. | Number of digits for display of biomarker data | 65 |
| 11.9. | Appendix | 9: Abbreviations & Trademarks | 66 |
| | 11.9.1. | Abbreviations | 66 |
| | 11.9.2. | Trademarks | 68 |
| 11.10. | Appendix | (10: List of Data Displays | 68 |
| | 11.10.1. | | 68 |
| | 11.10.2. | Mock Example Shell Referencing | 68 |
| | 11.10.3. | Deliverable [Priority] | 69 |
| | 11.10.4. | Study Population Tables | 70 |
| | 11.10.5. | Safety Tables | 73 |
| | 11.10.6. | Safety Figures. | 76 |
| | 11.10.7. | Efficacy Tables | 77 |
| | 11.10.8. | Efficacy Figures | 80 |
| | 11.10.9. | Pharmacodynamic Tables | 82 |
| | 11.10.10 | .Pharmacodynamic Figures | 83 |
| | 11.10.11 | .Biomarker Tables | 84 |
| | 11.10.12 | Biomarker Figures | 85 |
| | 11.10.13 | .Pharmacokinetic Tables | 86 |
| | | Pharmacokinetic Figures | 87 |
| | 11.10.15 | ICH Listings | 88 |
| | 11.10.16 | Non-ICH Listings | 93 |
| 11.11. | Appendix | 11: Example Mock Shells for Data Displays | 99 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| included in the Cili | iicai Study Ke | eport for Protocor. | | |
|---|---|---|---|---|
| Revision Chronology: | | | | |
| 2011N129686_00 | 2013-SEP-05 | Original | | |
| 2011N129686_01 | 2014-FEB-27 | Amendment N | No. 1 | |
| personnel; endpoin outpatient visits; en procedures; clarific removal of TCR cochange of volume r syringe, and removand Events Tables: outpatient visits; ad collected in additio 6.2.2); addition of I which ECGs will b months to Biomark to the first dose of shipped within 3 w 240mg/dL during 1 | t in table updated adpoint of glucation of time emplexes and required to pural of "micoportal fication of Day of the C-peptide ECGs at 6 house triplicate or the terms of the triplicate of triplicate of the triplicate of triplicate of the triplicate of the triplicate of the triplicate of triplicate of triplicate of the triplicate of tripli | ated to include instances added when period for collecting clarification of CE rege the IV infusion ore" from description that insulin should to 6 to footnote 18; are during the hypergurs post start of infusingle measures; ale; clarification that c-petion; clarification | summarising blinding status of ulin measurement for 7 days before performing MMTT and clamping information in the screening per D3 requirements throughout proton line and total volume filled into ion; the following changes to the T8 be recorded for 7 days before all clarification that glucose will be a glycaemic clamp procedure (Sect fusion (Section 6.2.3) clarification addition of TCR deep sequencing at MMTT will be at least 7 days peoptide and glucose samples will be that the hyperglycaemic range of the blood sampling time points. Amendment No. 2 | eriod; col; Time ion of at 24 prior pe |
| 2011N129686_02 | 20 | 014-APR-02 | Amendment No. 2 | |
| Hyperglycaemic events is included in the follow up endpoints and the Time and Events table to be consistent with the applicable secondary objective; rephrased "Immuno-Assay for syphilis test" in order to allow for different types of tests; increased the overage volume required to remain in the syringe for infusion; clarified the start of AE recording. | | | | Assay |
| 2011N129686_03 | 20 | 014-JUN-18 | Amendment No. 3 | |
| The third medical monitor has changed, therefore contact information for the replacement is included. The eligibility inclusion criterion was changed from two to one positive autoantibody associated with TIDM. | | | | |
| 2011N129686_04 | 20 | 014-JUL-28 | Republishing-Amendn<br>No. 3 | nent |
| | Clarified that within each cohort administration of study treatment for the first three patients will be staggered by at least three days across each centre. | | | |
| 2011N129686_05 | 20 | 015-FEB-11 | Amendment No. 4 | |

To increase flexibility for patients, dosing on Day 4, 5 & 6 may be performed on an outpatient basis if the Investigator is satisfied with the clinical status of the patient; clarification that if the infusion needs to be reduced or temporarily stopped the Investigator should first consult with the Medical Monitor who will consult the Sponsor, unless there is an immediate safety hazard, in this case the Investigator can inform the

Medical Monitor afterwards; clarified that insulin use is to be recorded prior to each visit and phone call; clarification that the decision to replace a patient is to be based on the reason for withdrawal; inclusion criteria # 3 amended; screen failure data are to be collected; assessments following patient withdrawal clarified; clarified that infusion kits are supplied to sites; assessment of EBV reactivation now conducted at 6 weeks after the first active dose (reduced from 12 weeks); blinding status amended to clarify that only the patient is blinded and not site staff; requirement for pharmacy staff to document that investigational product shipping conditions were 2-8°C included; anti-emetic added as a permitted concomitant medication, window of  $\pm 1$  day added to Day 14 and 21 visits and Week 4 telephone call; Section 6.2.2 amended to include a phone call at Week 4 to discuss AEs with patient and addition of assessments at Week 6; endpoints amended to reflect the change to visits at Week 4 and Week 6; Section 6.2.3 amended to include ECG at 3 hours and to clarify that assessments may stop at 3 hours post dose; clarification of cytokine release syndrome adverse events grading system and stopping criteria in Section 7.1.5; clarification on requirements for bilirubin samples included; CRO responsibilities clarified and supply of Ensure powder by CRO/GSK included.

| 2011N129686_06 | 2015-AUG-18 | Amendment No. 5 |
|----------------|-------------|-----------------|
|----------------|-------------|-----------------|

The assay for screening EBV IgG and IgM assessment was clarified in exclusion criterion number 18 and in Table 2 in the Risk Management section; exclusion criterion 18 was split into two exclusion criteria (18 and 19) to clarify EBV IgM, IgG and Viral load requirements for the interpretation of the results: a footnote was added to Table 6 (Stopping Criteria for CRS-Adverse Events) to provide further clarification regarding when individual stopping criteria are met; the dose preparation section was updated to clarify that an additional maximum of 30 minutes is allowed for dose preparation tasks and that if 6 hours is exceeded, the syringe and infusion materials must be replaced; EBV serology samples to assess IgG and IgM included for Day -1 in the Time and Events Table (Table 6.2.2 Dosing and Follow-Up).

Clarifications were made to the exploratory biomarker objectives and endpoints. Significant changes were: the addition of Th17 cells to the objective to assess the effect of otelixizumab on circulating lymphocytes; the addition of viral antigens to the endpoints to assess the effect of otelixizumab on the frequency of cytokine-producing antigen specific T cells; the addition of transcriptomic gene expression changes to the objective to assess the effect of otelixizumab on the clonal repertoire of circulating T cell populations; and clarification that the suppression activity of circulating T lymphocytes may be further evaluated by adapting assay conditions, possibly through adding and/or blocking of stimuli.

The Time and Events table was updated to show requirement for telephone calls at Month 36, 48 and 60.

Month 24 exploratory biomarkers are now being routinely collected and are not subject to the results of Month 12 biomarker analysis. In addition, it was clarified that Month 24 exploratory biomarker samples will be collected and only analysed after review of safety endpoints from Month 12 and not efficacy endpoints as previously stated.

Minor clarifications related to the Month 12 Interim Analyses were included.

| The name Quest was amende changed to Study Reference | ed to $Q^2$ Solutions and Study Pro<br>Manual. | ocedures Manual was |
|---|---|---|
| 2011N129686_08 | 2017-SEP-11 | Amendment No. 7 |
| removed from the Mixed Me<br>because the manufacturer (A | tly used Ensure powder (Abbot al Tolerance Test (Appendix 5) bbott) has discontinued the currefferent formulation. The details Reference Manual. | This has been amended rently used powder and the |
| 2011N129686_09 | YYYY-MMM-DD | Amendment No. 8 |

Data which emerged from an interim analysis carried out in this study showed a prompt regain of immune competence observed in treated subjects and consequent rapid resolution of EBV reactivation, both clinically and virologically. The long term EBV related PTLD risk, as observed in solid organ transplant on a chronic immune suppression therapy, is negligible.

Therefore, all references to month 48 and 60 have been removed as no patient currently enrolled in the study has reached month 48 of follow up. For the patients who have yet to complete their 24 month visit, this visit will be treated as a final visit and for those who have gone past month 24, they will be followed up with a final communication or visit (final follow up) upon approval of this protocol amendment.

Data from the literature identified a causal relationship between the degree of immunosuppression and an increased incidence of EBV related Post Transplant Lymphoprolerative Disorders (PTLD) and for this reason a long-term follow-up was implemented at the start of the study.

#### 1.1. RAP Amendments

Revision chronology:

| RAP Section | Amendment Details |
|---|---|
| Interim Reporting and Ar | nalysis plan OTX116505 [08-Dec-2014] |
| Reporting and analysis F 2.2, 2.3 | Plan OTX116505 Amend 1 [30-Sep-2015] Study objectives, endpoints and design updated to reflect protocol |
| • 4 | <ul> <li>amendment 5.</li> <li>Added in a 'Fully treated' population for use in key efficacy endpoints.</li> </ul> |
| • 6.2 | <ul> <li>Inclusion of a listing of concomitant medication during the dose escalations.</li> </ul> |
| • 7.1.2.1 | <ul> <li>Inclusion of additional safety outputs during the dose escalations.</li> </ul> |
| • 8.2.2.1 | <ul> <li>Additional sentence explaining the use of 'Fully Treated' population for Key<br/>efficacy outputs.</li> </ul> |
| • 11.2.3 | <ul> <li>Updated time and events table based on protocol amendment 5.</li> </ul> |
| • 11.2.4 | Updated time and events table based on protocol amendment 5. |

| RAP Section | Amendment Details |
|---|---|
| • 11.3 | <ul> <li>Baseline information added for antibody endpoints. RTF files will be produced<br/>for displays.</li> </ul> |
| • 11.4.2 | <ul> <li>Explanation of the derivation of a positive/negative value for the EBV IGm/IGg<br/>endpoint added</li> </ul> |
| • 11.5.1 | <ul> <li>Sentence added explaining that data after a subject withdraws will be listed<br/>and flagged</li> </ul> |
| • 11.5.3 | Explanation regarding handling of partial dates added. |
| • 11.6 | Update to PCI ranges |
| • 11.9 | <ul> <li>Inclusion of additional outputs as explained in sections 6.2, 7.1.2.1 and 8.2.2.1</li> </ul> |
| • 2.2 | <ul> <li>Exploratory Endpoints updated to reflect changes to protocol amendment<br/>dated 12SEP2016</li> </ul> |
| <ul><li>2.1</li><li>2.2</li></ul> | |
| • 3.1 | the exception of the second control of the s |
| | <ul> <li>Updated Interim analysis specifications to reflect changes to protocol</li> </ul> |
| | <ul> <li>Updated Interim analysis specifications to reflect changes to protocol<br/>amendment dated 12SEP2016</li> </ul> |
| ST-04457504 | <ul> <li>amendment dated 12SEP2016</li> <li>Clarification to process for delivering tables</li> </ul> |
| • 4 | amendment dated 12SEP2016 Clarification to process for delivering tables Biomarker endpoints added to ITT |
| | <ul> <li>amendment dated 12SEP2016</li> <li>Clarification to process for delivering tables</li> </ul> |
| • 4 | amendment dated 12SEP2016 Clarification to process for delivering tables Biomarker endpoints added to ITT |
| | amendment dated 12SEP2016 Clarification to process for delivering tables Biomarker endpoints added to ITT HLA-A2 Positive Population added |
| • 9 | amendment dated 12SEP2016 Clarification to process for delivering tables Biomarker endpoints added to ITT HLA-A2 Positive Population added New section to describe Exploratory Biomarker analysis |
| <ul><li>9</li><li>Appendix 8</li></ul> | amendment dated 12SEP2016 Clarification to process for delivering tables Biomarker endpoints added to ITT HLA-A2 Positive Population added New section to describe Exploratory Biomarker analysis New section to describe Exploratory Biomarker analysis Clarification to Laboratory parameters |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment dated on the 26 Oct 2017 for the study GSK2136525/OTX116505 (GSK Document No.: 2011N129686 09).

# 2.2. Study Objective(s) and Endpoint(s)

| Primary | |
|---|---|
| Primary Objectives (Safety) | Primary Endpoints (Safety) |
| To assess the effect of a single course of otelixizumab treatment on the acute and long term safety and tolerability of otelixizumab in NOT1DM patients. | <ul> <li>Incidence of adverse events (AEs) particularly those related to Cytokine release syndrome (CRS).</li> <li>Epstein-Barr virus (EBV) reactivation over Day 21 to Month 24.</li> <li>Changes in laboratory values, electrocardiograms (ECGs) and vital signs over Day 14 to Month 24.</li> </ul> |

| Secondary Secondary Objectives (Pharmacokinetic) | Secondary Endpoints (Pharmacokinetic) |
|---|---|
| To assess the pharmacokinetics of repeat<br>dose administration of otelixizumab over 14<br>days in NOT1DM patients. | Free serum otelixizumab concentrations over<br>Days 1-14 and summary PK parameters. |
| Secondary Objectives (Efficacy) | Secondary Endpoints (Efficacy) |
| <ul> <li>To assess the effect of a single course of<br/>otelixizumab treatment on the rate of decline<br/>of pancreatic β-cell function over 24 months in<br/>NOT1DM patients.</li> </ul> | Change from baseline in C-peptide and glucose AUC (0-120) after a Mixed Meal Tolerance Test at Month 3, 6, 12, 18 and 24. |
| <ul> <li>To assess the effect of a single course of<br/>otelixizumab treatment on the rate of decline<br/>of C-peptide response and insulin sensitivity of<br/>β-cell function determined after a<br/>hyperglycemic clamp over 24 months in<br/>NOT1DM patients.</li> </ul> | Change from baseline in C-Peptide and glucose AUC hyperglycemic phase [H60 to H140 minutes] and insulin sensitivity (IS) index after a hyperglycemic clamp at Months 6 and 24. |
| <ul> <li>To assess the effect of a single course of<br/>otelixizumab treatment on exogenous insulin<br/>use for otelixizumab over 24 months in<br/>NOT1DM patients.</li> </ul> | Change from baseline in mean daily insulin<br>use over 7 consecutive days during the week<br>preceding all visits and phone calls. |
| To assess the effect of a single course of otelixizumab treatment on glycaemic control over 24 months in NOT1DM patients. | <ul> <li>Change from baseline in HbA1c level.</li> <li>Body weight Day -1, Months 12-24.</li> <li>Hypoglycemic &amp; hyperglycemic events over<br/>Months 1-24.</li> </ul> |
| Secondary Objectives (Pharmacodynamic) | Secondary Endpoints (Pharmacodynamic) |
| <ul> <li>To assess the effect of a single course of<br/>otelixizumab treatment on the time course and<br/>magnitude of CD4+ and CD8+ cells and CD3<br/>binding and saturation on all these cells during<br/>repeat dose administration of otelixizumab</li> </ul> | Relative change from baseline (%) in CD4+<br>and CD8+ cells, free CD3 and bound<br>otelixizumab on CD4+ and CD8+ cells on<br>Days 1 through 14. |

| over 14 days in NOT1DM patients. | |
|---|---|
| To assess the effect of a single course of otelixizumab treatment on the immunogenicity of otelixizumab in NOT1DM patients. | <ul> <li>Change from baseline in anti-drug antibody<br/>levels at Months 3 and 6.</li> </ul> |
| Exploratory Objectives * | Exploratory Endpoints * |
| To assess the effect of a single course of otelixizumab treatment on circulating lymphocyte populations over 24 months in NOT1DM patients. | <ul> <li>Change from baseline in absolute lymphocyte<br/>counts and ratios in some or all, but not<br/>limited to subsets (CD3+ CD4+, CD3+ CD8+,<br/>and CD19+ cells) and phenotype (e.g.<br/>effector, memory, regulatory T cells, e.g.<br/>CD45RA, CCR7+) over Week 6 to Month 24.</li> </ul> |
| To assess the effect of a single course of otelixizumab treatment on circulating lymphocutes such as regulatory T cell numbers (as quantified by CD3 and demethylated FoxP3 expression) and Th17 cells over 24 months in NOT1DM patients. | <ul> <li>Change from baseline in cell-type specific<br/>methylation marker expression in some or all,<br/>but not limited to CD3, FoxP3 and Th17 in<br/>whole blood over Week 6 to Month 24.</li> </ul> |
| To assess the effect of a single course of otelixizumab treatment on absolute numbers and ratios of circulating antigen specific CD8+ T cells over 24 months in HLA-A2+ NOT1DM patients. | <ul> <li>Change from baseline in absolute numbers<br/>and ratios of HLA-A2-restricted CD8 T<br/>lymphocytes reactive to specific auto-antigens<br/>(by multimer) over Week 6 to Month 24.</li> </ul> |
| To assess the effect of a single course of otelixizumab treatment on frequency of cytokine-producing antigen specific T cells over 24 months in NOT1DM patients. | <ul> <li>Change from baseline in frequency of<br/>cytokine producing cells following in vitro<br/>stimulation with auto-antigens and viral<br/>antigens (by ELISPOT) over Week 6 to<br/>Month 24.</li> </ul> |
| To assess the effect of a single course of otelixizumab treatment on serum auto-antibodies titers and serum analytes associated with treatment or autoimmune pathology over 24 months in NOT1DM patients. | <ul> <li>Change from baseline in auto-antibody titres<br/>(using a panel of common auto-antibodies<br/>associated with T1DM antigens and possibly<br/>other auto-antigens) and serum analytes<br/>(such as cytokines/ chemokines) during the<br/>first 14 days of treatment and over Week 6 to<br/>Month 24.</li> </ul> |
| To assess the effect of a single course of otelixizumab treatment on clonal repertoire of circulating T cell populations and/or transcriptomic gene expression changes over 24 months in NOT1DM patients. | <ul> <li>Change from baseline in T cell clonal repertoire by TCR deep sequencing over Day 6 to Month 24.</li> <li>Change from baseline in transcriptomic gene expression profile(s) by micro-array and/or alternative equivalent technologies including RNA sequencing at selected timepoint(s) post dosing.</li> </ul> |
| <ul> <li>To assess the effect of a single course of<br/>otelixizumab treatment on β-cell death over<br/>24 months in NOT1DM patients.</li> </ul> | <ul> <li>Change from baseline in serum by measuring<br/>relative levels of unmethylated INS DNA<br/>and/or other biomarkers for β-cell death in<br/>serum over Week 6 to Month 24.</li> </ul> |
| To assess the effect of a single course of otelixizumab treatment on suppression activity of circulating T lymphocytes over 24 months in NOT1DM patients. | <ul> <li>Change from baseline in relative levels of T<br/>lymphocyte suppression using micro<br/>suppression assay over Week 6 to Month 24.</li> <li>Suppression activity may be further evaluated<br/>by adapting assay conditions possibly through<br/>adding and/or blocking of stimuli.</li> </ul> |

| <ul> <li>To assess long term safety follow-up with otelixizumab treatment.</li> <li>Severe (as per ADA classification, Protocol Appendix 7) hypoglycemic events which occurred following Month 24 visit (if available) until final follow-up</li> <li>Severe hyperglycemic events which occurred following Month 24 visit (if available) until final follow-up</li> <li>Mean daily insulin use over 7 consecutive days preceding the call.</li> <li>HbA1c results around time of the phone call.</li> </ul> | Follow up Objectives | Follow up Endpoints |
|---|---|---|
| | [집] [지 : [지지] [집 : [지 : [대] [지 : [대] | <ul> <li>Severe (as per ADA classification, Protocol Appendix 7) hypoglycemic events which occurred following Month 24 visit (if available) until final follow-up</li> <li>Severe hyperglycemic events which occurred following Month 24 visit (if available) until final follow-up</li> <li>Mean daily insulin use over 7 consecutive days preceding the call.</li> </ul> |

# 2.3. Study Design



Note: the study design shown is the original study design. Stopping criteria for escalation was met in Cohort 3. In addition, the duration of the study has been shortened to 24 months.

| Cohort 3. In addition, the duration of the study has been shortened to 24 months. | |
|---|---|
| Overview of Key Study | y Design Features |
| Design Features | <ul> <li>Multi-centre, single-blind, randomised, placebo-controlled 6 day repeat<br/>dose study to investigate the safety, tolerability, pharmacokinetics,<br/>pharmacodynamics, efficacy &amp; immunological profile of intravenously<br/>administered otelixizumab in New Onset Type 1 Diabetes Mellitus<br/>(NOT1DM) patients.</li> </ul> |
| Dosing | <ul> <li>Patients dosed within ~ 28 days of diagnosis (not more than 32 days).</li> <li>Insulin usage documented for ~ 7 days prior to screening &amp; Day -1 (baseline).</li> <li>There will be a 7-21 day period from screening to admission to the clinic on Day -2 for the first overnight stay of the in-patient period.</li> <li>Patients randomised on Day -1 followed by a hyperglycaemic clamp test.</li> <li>Dosing will start on Day 1 &amp; patients will remain in unit for IV dosing.</li> <li>Patients will be given the following flexible options for dosing on Days 4, 5 and 6: Option 1: Receive study treatment on an out-patient basis on any of Days 4, 5 or 6, if the Investigator is satisfied with the clinical condition of the patient. Option 2: Patients will remain in the unit if there are any concerns about their clinical status, or if the patient prefers to remain in the unit for logistical reasons.</li> <li>NOTE: Within each cohort administration of study treatment will be staggered by at least three days for the first three patients across each centre.</li> </ul> |
| Treatment<br>Assignment | <ul> <li>Approximately 32 patients will be dosed in a dose escalation design exploring 4 dose cohorts (4 dose levels (9, 18, 27,36) and placebo).</li> <li>At each dose cohort 8 patients will be randomised to otelixizumab and 2 patients to placebo.</li> </ul> |
| Interim Analysis | The planned protocol defined unblinded interim analyses were: |

| 0 0 | Ongoing data reviews throughout the trial progression. Data reviews to assess whether to dose escalate to the next cohort. |
|---|---|
| 0 | 12 months formal interim analysis. |

# 2.4. Statistical Hypotheses

The protocol defined hypotheses were defined as:

- As the primary objective is to assess the safety, tolerability and maximum tolerated dose of Otelixizumab in participants with NOT1DM patients, there are no formal hypotheses being tested in the study; instead an estimation and inference approach will be adopted to evaluate the objectives.
- If data permits, a model-based approach will be used to characterise and assess any
  evidence of dose response relationships with endpoints of interest.

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

The interim analyses are described in the interim RAP, Amendment 2, dated 01-Nov-2016 and include the following.

| Interim<br>Analysis | Details (Protocol Defined) |
|---|---|
| During The<br>Study | <ul> <li>There will be ongoing data reviews conducted by the study team of the unblinde<br/>safety and efficacy data, and any available pharmacokinetic and<br/>pharmacodynamic data throughout the trial progression.</li> </ul> |
| Dose<br>Escalation | Further unblinded data reviews of safety data will be performed to support whether to dose escalate to the next cohort. If deemed appropriate, the review may also include supportive pharmacokinetic, biomarker or pharmacodynamic data if available. Details are provided below: |
| | <ul> <li>Data will be reviewed after 10 patients have been dosed in cohort 1 (8 patients on otelixizumab 9 mg and 2 patients on placebo) and have completed approximately 6 wks of the study and required data is available.</li> </ul> |
| | <ul> <li>If required, data reviews prior to 6 wks may also be conducted to facilitate<br/>dose escalation to the next cohort.</li> </ul> |
| | <ul> <li>It is not expected that this review will occur on fully cleaned data.</li> </ul> |
| | <ul> <li>Further data reviews based on criteria provided for cohort 1, will be performed<br/>for subsequent cohorts, including an overall review of accumulated data<br/>across the cohorts.</li> </ul> |
| | <ul> <li>Core members of the dose escalation review team will include the principal<br/>investigator (Chief), medical monitor, GCSP, clinical pharmacologist, study<br/>leader &amp; statistician. Other GSK and CRO study team members may be</li> </ul> |

| Interim<br>Analysis | Details (Protocol Defined) |
|---|---|
| | included as required. |
| 12 Months | <ul> <li>A formal unblinded interim analysis is also planned to occur.</li> <li>The first interim will occur when all patients in cohorts 1 and 2 have completed 12 months study duration, but may also include any available data from subsequent cohorts 3 and 4 as appropriate.</li> </ul> |
| | <ul> <li>The second interim analysis will occur when all patients from the last fully<br/>enrolled cohort (i.e. not stopped due to safety / tolerability) have completed 12<br/>months study duration. The purpose of this interim analysis is to provide the<br/>project team and GSK stakeholders with key data to inform internal decision<br/>making, in order to plan future studies within the clinical development for the<br/>asset.</li> </ul> |
| | There are no planned implications for the conduct of the study. |
| | <ul> <li>Appropriate data summaries will be at the treatment group level for key endpoints of interest and the circulation of results will be restricted to selected members of the project team and key GSK stakeholders. Results or discussions will not be circulated to blinded staff involved in the conduct of the study at the sites.</li> </ul> |
| | Note: Because of the anticipated time frame to process and analyse the biomarker data they will not be included in the SAC deliverables. Therefore all other data may be frozen and the study unblinded before they are available. Once the data become available they will be added to the other frozen datasets and analysed as described |

# 3.2. Final Analyses

The following final planned analyses will be performed and details will be provided in this RAP.

| Analysis | Details |
|---|---|
| Final Primary Analyses<br>(24 Months) | The final analysis will occur when the last planned cohort (i.e. based on the dose escalation criteria) have completed 24 months study duration or have had a final follow-up for subjects who, at the time of the implementation of Amendment 08 of the protocol, will have already reached months 24. |

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|-------------|-----------------------|-------------------------|
| 1 opulation | Dominion / Ontona | Litapoliti(o) Evaluated |

| Population | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|
| Screened<br>Population | All participants who were screened for eligibility | <ul><li>Study Population</li><li>Screening Failures</li></ul> |
| Randomized<br>Population | <ul> <li>All participants who were randomly assigned to a study treatment</li> <li>In summary tables, the treatment the subject was randomized to will be used</li> </ul> | Study Population |
| Enrolled<br>Population | <ul> <li>All participants who passed screening, signed informed consent and entered the study. This includes: <ul> <li>Run-in failures</li> <li>Randomised participants</li> </ul> </li> <li>Screening failures are not included</li> </ul> | Assignment to Analysis Populations |
| Safety<br>Population | <ul> <li>Comprise of participants who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment which the participant actually received.</li> </ul> | <ul><li>Study Population</li><li>Safety</li><li>Pharmacodynamic</li></ul> |
| Intent-To-<br>Treat<br>(Treated) | <ul> <li>Comprise of all randomised participants who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment to which the participant was randomised.</li> </ul> | Efficacy Biomarker |
| Per-Protocol<br>Population<br>(Treated) | <ul> <li>Comprise of all randomized participants who receive at least one dose of study treatment and who comply with the protocol.</li> <li>Protocol deviations that would exclude participants from the PP population are defined in the Protocol Deviation Management Plan (PDMP) Version 2.5, dated 25-Jul-2018. If the PDMP is updated after signature of the SAP and before database lock, then the newest version will be used instead.</li> </ul> | As required based on data and exclusion of participants. |
| Fully treated | Comprise of all randomized participants who receive the full 6 days of treatment based on actual exposure data. | <ul> <li>Population may<br/>also be used for<br/>the key efficacy<br/>endpoints</li> <li>Population may be<br/>used for PK and<br/>biomarker<br/>analyses</li> </ul> |
| Multimer<br>Analyses<br>Population | Comprises of all Intent-to-treat (Treated) who have available multimer data | Biomarker (Multimer Analysis) |

| Po | pulation | Definition / Criteria | Endpoint(s) Evaluated |
|---|---|---|---|
| • | Please refe | r to Appendix 10: List of Data Displays, which details the p | opulation for each display generated. |

- to the state of th
- As there are no planned pharmacokinetic analyses, this population will be defined for the next reporting effort.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study according to the Protocol Deviation Management Plan. Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorized on the protocol deviations dataset. This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion form.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Study Treatment Descriptions | | |
|---|---|---|---|
| Code | Code Description Description | | |
| Α | Otelixizumab 9 mg | OTX 9 mg | 2 |
| В | Otelixizumab 18 mg | OTX 18 mg | 3 |
| С | Otelixizumab 27 mg | OTX 27 mg | 4 |
| P [1] | Placebo | Placebo | 1 |

#### NOTES:

- [1] Placebo will be pooled across cohorts for analysis and reporting.
- [2] Order in which treatments are to be presented in Tables, Figures and Listings.

Due to protocol amendments, there have been some changes in the scheduling of certain assessments. Listings will show the visit according to the schedule according to the protocol version used, while for summary tables the following rules shall apply:

- In general, if for an endpoint some participants have a Week 4 assessment, while other subjects have a Month 1 assessment (e.g. mean insulin usage), it will be summarized under Week 4.
- For vital signs, haematology, clinical chemistry, biomarkers and Epstein-Barr virus serology, the time points Month 1 and Week 6 shall be combined and displayed as "Month 1/Week 6" with an explanatory footnote.

Treatment comparisons will be displayed as follows using the descriptors as specified:

- 1. OTX 9 mg vs Placebo
- OTX 18 mg vs Placebo
- 3. OTX 27 mg vs Placebo

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

As triplicates are taken for the baseline ECG data, the average will be used as baseline. If one or two of the triplicate measurements are missing, the remainding measurement(s) will be used to calculate the average. For categorical variables for triplicate ECG assessments the worst case will be used. In terms of worseness this is defined as abnormal, clinically significant > abnormal, clinically insignificant > normal > unable to evaluate.

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Table 1 provides an overview of appendices within the final RAP for outlining general considerations for data analyses and data handling conventions.

- There are planned examination of covariates and subgroups.
- There are no planned adjustments made for multiple centres in this study.
- There are no planned adjustments for multiple comparisons or multiplicity.
- There are known discrepancies between the terminology subject vs participant used across Protocols and RAP. All displays will use the term 'Subjects'.
- In the following the use of the word "log" is to be understood to refer to the natural logarithm (base e) unless another base is specifically stated

#### Table 1 Overview of Appendices

| Section | Component |
|--------------|--------------------------------------------------------------|
| 11.1 | Appendix 1: Schedule of Activities |
| <b>1</b> 1.2 | Appendix 2 Assessment Windows |
| 11.3 | Appendix 3: Study Phases |
| 11.4 | Appendix 4: Data Display Standards & Handling Conventions |
| <b>1</b> 1.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |
| 11.8 | Appendix 8: Biomarker Analyses |
| 11.9 | Appendix 9: Abbreviations & Trademarks |
| 11.10 | Appendix 10: List of Data Displays |
| 11.11 | Appendix 11: Example Mock Shells for Data Displays |

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the Enrolled population, unless otherwise specified.

Study population analyses including analyses of participants disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards.

Full details of data displays being presented in Appendix 10: List of Data Displays.

## 6.2. Exposure

Cumulative dose, days on study drug and daily infusion duration in hours for each dosing day will be summarised.

# 6.3. Concomitant Medication and Insulin Usage

All concomitant medication will be summarised and listed as per GSK Core Data Standards. To aid review of concomitant medications, the data collected for the daily insulin use will be listed separately.

## 7. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified. Due to the long duration of the study safety summaries will be presented for the following time spans: Overall, Dosing Period (defined as day of first dose up to and including day of last received dose of study drug), Post dose up to Week 6, Post-Week 6. A definition is found in Section 11.3.

# 7.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 10: List of Data Displays.

No separate outputs will generated for Common AEs (more than 5% incidence in any treatment group) as the sample size means all occurrences would be considered common. A footnote will be added to the all AE overview, that all categories count as common.

In case of liver monitoring/stopping events, the outputs required by GSK guidelines will be produced. Those output are not listed in Section 11.10.

#### 7.2. Adverse Events Related to CRS and EBV Reactivation

Adverse Events associated with Cytokine Release Syndrome (CRS) induced symptoms and events associated with EBV reactivation will be summarised as per section 7.1 as well as summarised in separate outputs.

See Section 11.5.3 for details on selection of AEs related to CRS and EBV reactivation. The details of the planned displays are provided in Section 11.10. List of Data Displays.

# 7.3. EBV Serology and Viral Load

EBV Serology will be listed and summarised using frequency of positive/negative values at each visit as described in Section 11.5.3

EBV Viral Load will be listed and summarised using summary statistics using a log-10 transformation. Frequency of number of copies per 10^6PBM Cells will presented as described in Section 11.5.3.

#### 7.4. Cardiovascular Events

Event Specific data will be listed if there are any occurences of cardiovascular events. If there are no events these listings will not be produced.

# 7.5. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Section 11.10.

# 7.6. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Section [11.10]: List of Data Displays.

#### 8. PHARMACOKINETIC ANALYSES

#### 8.1.1. Drug Concentration Measures

Blood sampling time will be related to the start of dosing. Linear and semi-logarithmic individual serum concentration-time profiles and mean (±SD) and median profiles will be plotted by treatment.

Serum concentrations of otelixizumab will be listed and summarised by treatment group and nominal time.

Refer to Section 11.4 for the reporting process and standards.

## 8.2. Derived Serum Pharmacokinetic Parameters

- Free serum otelixizumab pharmacokinetic parameters will be calculated using SAS.
   Calculations will be based on the actual sampling times recorded during the study.
- From the serum concentration-time data, the pharmacokinetic parameters in Table 2 will be determined for free serum otelixizumab, as data permit, for each treatment and for each participant.

#### • Table 2 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed serum concentration |
| tmax | Time to Cmax |
| AUC(0-τ) | Area under the serum concentration-time curve from time zero over the dose interval |

NOTES: Additional parameters may be included as required.

 $AUC(0-\tau)$  will be calculated using the trapezoidal rule (see section 11.5.4) and will use all timepoints up to and including Day 6, 1 hour post dose.

## 9. EFFICACY ANALYSES

# 9.1. Overview of Planned Efficacy Analyses

Following review of the data, additional analyses may be conducted to further support the evaluation and interpretation of the data. Details of data displays being presented in Section 11.10: List of Data Displays.

# 9.1.1. Endpoints / Variables

The following endpoints will be analysed:

- Change from Baseline in Weighted Mean AUC (0-120) C-Peptide & Glucose from MMTT
- Change from Baseline in Weighted Mean AUC [(60-140)] C-Peptide & Glucose from Hyperglycemic Clamp Test
- Change from Baseline in Insulin Sensitivity Index from Hyperglycemic Clamp Test
- Change from Baseline in Mean Daily Insulin Use
- Change from Baseline in %HbA1c
- Change from Baseline in Body Weight
- Hypoglycemic and hyperglycemic events over Months 1-24.
- Number (percent) of participants meeting responder status on C-peptide from MMTT
- Number (percent) of participants achieving partial remission status
- Number (percent) of participants achieving HbA1c Responder Status

For detailed derivations of the efficacy endpoints please see Section 11.5.4.

# 9.1.2. Summary Measure

For continuous measures the treatment comparison will be the difference between treatment means at each visit. If log transformation is required the treatment comparison will be the ratio of treatment means at each visit.

For responder endpoints the treatment comparison will be the difference in % of responders in each treatment group.

#### 9.1.3. Population of Interest

The efficacy analyses will be based on the Intent-To-Treat (Treated) population, unless otherwise specified.

## 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

No imputation of missing data will be performed.

# 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Section 11.10: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

Responder endpoints will be summarised only.

#### 9.1.5.1. Statistical Methodology Specification - MMRM

#### **Endpoints**

- Change from Baseline in Weighted Mean AUC (0-120) C-Peptide & Glucose from MMTT
- Change from Baseline in Weighted Mean AUC [(60-140)] C-Peptide & Glucose from Hyperglycemic Clamp Test
- Change from Baseline in Insulin Sensitivity Index from Hyperglycemic Clamp Test
- Change from Baseline in Mean Daily Insulin Use
- Change from Baseline in %HbA1c
- Change from Baseline in Body Weight

#### **Model Specification**

 Endpoints will be statistically analysed using a mixed model repeated measures (MMRM) model.

Terms fitted in the MMRM model will include:

- Fixed Categorical: Treatment, Visit, Treatment \* Visit Interaction
- Fixed Continuous Covariates: Baseline #
- Repeated: Visit

Other covariates may be added using the following procedure:

For each covariate the MMRM model for the MMTT C-peptide analysis using the ITT population will be expanded and fitted two times:

- Only the covariate will be added as an additional fixed factor
- Both the covariate and the interaction of the covariate with treatment will be added as fixed factors

If the covariate is significant at a 10% alpha level using Type III p-values in the first model, then the covariate may be added to all MMRM models of efficacy endpoints or specific analyses may be repeated with the covariate added. When the interaction between the covariate and treatment is significant at a 10% alpha level in the second model, then both the covariate and the interaction of the covariate with treatment may be added.

The following covariates will be considered: BMI, Weight, Number of positive Auto Antibodies (categorical, 1 or > 1; see Section 11.5.3 for derivation).

The p-values for the tests described above will be presented in the statistical listing for the MMTT C-peptide analysis.

## **Model Checking Assumptions**

- Model assumptions will be applied, but appropriate adjustments may be applied based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
  - In the event that this model fails to converge, alternative correlation structures may be considered such as Spatial Power Model, CSH or CS. The correlation structure chosen should make sense and not just chosen because model converges (e.g. AR(1) would not be appropriate as the visit structure is not even).
  - Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.
- All model checking will be presented in a statistical listing along with the raw SAS output from the analyses.

#### Presentation of Results

- Adjusted means (Value and Change from Baseline) and corresponding standard error of means (SEs) and 95% confidence intervals will be presented for each treatment by time, together with estimated treatment differences and the corresponding 95% confidence intervals.
- Plots of LS means =/- SE from the model will be generated for each treatment by time.
   Additionally, plots of differences and 95% confidence intervals for the comparison of interest will be generated.

#### Sensitivity and Supportive Analyses

- A supportive analysis using the 'Fully Treated' population will be performed for the following endpoints:
  - Change from Baseline in Weighted Mean AUC (0-120) C-Peptide & Glucose from MMTT
  - Change from Baseline in Weighted Mean AUC (60-140) C-Peptide & Glucose from Hyperglycemic Clamp Test

# 9.2. Overview of Planned Pharmacodynamic Analyses

# 9.2.1. Endpoints / Variables

The following endpoints will be analysed:

• Relative change from baseline (%) in CD4+ and CD8+ cells, free CD3 and bound otelixizumab on CD4+ and CD8+ cells on Days 1 through 14.

## 9.2.2. Summary Measure

The target engagement variables (see Section 11.5.5 for a detailed listing and derivations) will be summarized. The treatment comparison will be the difference between treatment means at each visit.

#### 9.2.3. Population of Interest

The pharmacodynamic analyses will be based on the Fully Treated Population unless otherwise specified. Listings will be created using the Safety Population.

## 9.2.4. Strategy for Intercurrent (Post-Randomization) Events

No imputation of missing data will be performed.

#### 9.2.5. Statistical Analyses / Methods

Analysis will be restricted to summary statistics. Details of the planned displays are provided in Section 11.10 List of Data Displays and will be based on GSK data standards and statistical principles.

## 9.3. Pharmacokinetic / Pharmacodynamic Analyses

No PK/PD Analyses are considered to be in the scope of this RAP.

# 9.4. Overview of Planned Exploratory Analyses

# 9.4.1. Endpoints / Variables

The following endpoints will be analysed as available:

- Frequency and phenotype of lymphocyte subsets by flow cytometry
- Frequency and phenotype of lymphocyte subsets by flow cytometry by C-peptide Responder Status
- Frequency and phenotype of HLA-A2-resticted T1D- and EBV-specific CD8+ T cells by multimer analysis
- Quantification of serum cytokines and soluble cytokine receptors
- Percentage Productive clonality by TCR deep sequencing

Due to data quality the remaining biomarker data will be listed only:

Details of data displays being presented in Section 11.10.

Further details of the endpoints to be considered is presented in Section 11.8.

# 9.4.2. Summary Measure

For continuous measures the treatment comparison will be the difference between treatment means at each visit. If log transformation is required the treatment comparison will be the ratio of treatment means at each visit.

## 9.4.3. Population of Interest

Figures will be based on the Fully Treated Population. For the other outputs the ITT Population will be used, with the exception of the multimer analysis, which will be performed using the Multimer Analyses Population.

## 9.4.4. Strategy for Intercurrent (Post-Randomization) Events

No imputation of missing data will be performed.

# 9.4.5. Statistical Analyses / Methods

Analysis will be restricted to summary statistics. Details of the planned displays are provided in Section 11.10: List of Data Displays and will be based on GSK data standards and statistical principles.

## 10. REFERENCES

- 1. GlaxoSmithKline Document Numbers 2011N129686\_00 (Original 05-Sept-13), 2011N129686\_01 (Protocol Amendment 27-Feb-14), 2011N129686\_02 (Protocol Amendment 02-APR-14), 2011N129686\_03 (Protocol Amendment 28-JUN-14), 2011N129686\_04 (Republish Protocol Amendment 28-JUL-14), 2011N129686\_05 (Protocol Amendment 11-FEB-15), 2011N129686\_06 (Protocol Amendment 18-AUG-15), 2011N129686\_07 (Protocol Amendment 12-SEP-16), 2011N129686\_08 (Protocol Amendment 11-SEP-17), 2011N129686\_09 (Protocol Amendment 26-OCT-17): A Single Blind, Randomised, Placebo Controlled, Repeat Dose, Dose Escalating Study Investigating Safety, tolerability Pharmacokinetics, Pharmacodynamics and the Beta-Cell Preserving Effect of Otelixizumab in New-Onset, Autoimmune Type 1 Diabetes Mellitus Patients.
- GlaxoSmithKline Interim Reporting and Analysis Plan OTX116505 (Original 08-Dec 2014), Interim Reporting and Analysis Plan OTX116505 Amendment 1 (30-Sep-2015), Interim Reporting and Analysis Plan OTX116505 Amendment 2 (01-Nov-2016).
- 3. Mortensen, H. B., et al. (2009). "New definition for the partial remission period in children and adolescents with type 1 diabetes." Diabetes Care 32(8): 1384-1390.
- 4. Long, S. A., et al. (2016). "Partial exhaustion of CD8 T cells and clinical response to teplizumab in new-onset type 1 diabetes." Sci Immunol 1(5).
- 5. DeFronzo, R. A. et al. (1979). "Glucose clamp technique: a method for quantifying insulin secretion and resistance." Am. J. Physiol. 237(3).

# 11. APPENDICES

# 11.1. Appendix 1: Schedule of Activities

# 11.1.1. Protocol Defined Time & Events

# 11.1.2. Screening

| Medication history |
|---|
| Full physical examination (including height and weight) |
| Drug/alcohol history |
| Chest X-ray (to rule out TB) |
| Serology (EBV, HIV, Hep C, Hep B, Syphillis) |
| 12-lead ECG in triplicate |
| Vital signs (including temperature, blood pressure and pulse rate (in triplicate) and respiration rate |
| Urine Pregnancy test (female only) |
| Haematology (must include total lymphocyte count) |
| Clinical Chemistry |
| T1DM Auto antibody (Anti-GAD, anti-IA2, antibody to islet cell antigen (ICA), anti-ZnT8) |
| EBV Viral Load (PCR) |
| AE assessment |

| The following must be performed at least 7 days prior to dosing |
|-----------------------------------------------------------------|
| Mixed Meal Stimulated C-peptide (MMTT) |

# 11.1.3. Dosing and Follow-Up

| | | | | | | Day | | | | | Month | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 14 | 21 | Week<br>4 | Week<br>6 | 2 | 3 | 6 | 9 | 12 | 18 | 24 | 36<br>month<br>(if<br>applicab<br>le)<br>and/or<br>final<br>follow<br>up |
| Patient admitted to unit <sup>1</sup> | Χ | | | | | | | | | | | | | | < | | | | | |
| In Patient | | Х | X | Х | Χ | X <sup>2</sup> | X <sup>2</sup> | X2 | | | | | | | | | | | | |
| Prophylaxis then IV Dosing of study treatment | | | Χ | Х | Х | Х | Х | Х | | | | | | | | | | | | |
| Patient Discharged <sup>2</sup> | | | | | | | | Х | | | | | | | s. | | | , | | |
| Out Patient# | | | | | | Х | Х | Х | Х | Х | | X | Χ | Х | Χ | X | Χ | Х | Χ | |
| Telephone call or out-patient visit to collect<br>AEs, hypoglycemic and hyperglycemic events<br>and concomitant<br>medication use | | | | | | | | | | | Х | | | | | | | | | Х |
| Brief Physical Examination | | Х | X3 | X3 | <b>X</b> 3 | X3 | <b>X</b> 3 | X3 | Х | Х | | X | Χ | Х | Χ | X | Χ | Х | Х | |
| 12 lead ECG <sup>4,6</sup> | | Х | Х | X | Х | Х | Х | Х | Х | | | | | | | | Χ | | Χ | |
| Vital Signs <sup>5,6</sup> | | Χ | Χ | X | Χ | Χ | Х | Χ | Х | Х | el. | Χ | Χ | Х | Χ | X | Χ | Χ | Χ | |
| Serum Pregnancy Test | | X | | | | | | | | | | X | Χ | Х | Χ | X | Χ | Χ | Χ | |
| Alcohol & drugs of abuse test | | Х | | | | | | | | | | | | | | | | | | |
| Haematology <sup>7</sup> | | Χ | | Х | Χ | Х | Х | Х | Х | Х | | Х | Χ | Х | Χ | X | Χ | Χ | Χ | |
| Clinical Chemistry <sup>7</sup> | | Χ | Χ | Х | Χ | Х | Х | X8 | Х | | | Х | | Х | Χ | X | Χ | Χ | Χ | |
| HSV-1 & HSV-2 IgG & IgM <sup>9</sup> | | Х | | | | | | | | | | | | | | | | | | |
| EBV Viral Load (PCR) <sup>7</sup> | | Χ | | | | | | Х | | Х | | Χ | Χ | Х | X10 | | | | Χ | |
| EBV Serology - IgG and IgM 7 | | Χ | | | | | | Х | | Χ | | Х | Χ | Х | Χ | | Χ | 0. 0 | Χ | |
| CMV Serology - IgG and IgM7 | | Х | | | | | | Х | | | | Χ | Χ | Х | Χ | | Χ | 4. | Х | |

| | | | | | 015 | Day | | | | | | | | 075 . 7 * | М | onth | ì | | 7 | 390 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | -2 | -1 | 1 | 2 | 3 | 4 | 5 | 6 | 14 | 21 | Week<br>4 | Week<br>6 | 2 | 3 | 6 | 9 | 12 | 18 | 24 | 36<br>month<br>(if<br>applical<br>le)<br>and/or<br>final<br>follow<br>up |
| PK Blood Sample <sup>6</sup> | | | Х | X | Х | Х | Х | Х | X11 | | | | | | | | | | | |
| CD3 Saturation, free CD3 bound otelixizumab<br>/CD4+/CD8+ Blood Sample <sup>6</sup> | | | х | Х | Х | Х | Х | Х | X11 | - | | | | | | | | | | |
| Record insulin usage for 7 days before visit / call | | Х | | | | | | | Х | Х | Х | Х | Х | х | Х | Х | Х | Х | Х | Х |
| AE Assessment | | | <> | | | | | | | | | | | | | | | | | |
| Concomitant Medication Review | | | < | | | | | | | | | | | | | | | | | > |
| Hypoglycaemic / Hyperglycaemic Events | | | < | | | | | | | | | | | | | | | | | > |
| Anti-GAD, anti-IA2, antibody to islet-cell antigen (ICA), anti-ZnT8 & Insulin-antibodies (IAA) | | Х | | | | | | | | | | | | | | | | | | |
| Anti-otelixizumab antibodies Blood Sample | | Χ | | | | | | | | 6 5 | | | | Х | Χ | | | | | |
| Mixed Meal Stimulated C-peptide (MMTT) <sup>12</sup> | | | | | | | | | | | | | | Х | X14 | | Χ | Х | X14 | |
| Beta Cell Function by Hyperglycaemic Clamp <sup>13</sup> | | Χ | | | | | | | | | | | | | X14 | | | | X14 | |
| HbA1c | | Χ | | | | | | | | | | | | | Х | | Χ | | Х | X15 |
| Bodyweight | | Х | | | | | | | | | | Х | Х | Х | Х | Х | Х | Х | Х | |
| Various Blood samples for Exploratory Biomarkers | | Х | | | | | | X16 | | | | Х | | X | Х | | Х | | X17 | |
| Saliva sample for Pharmacogenetics (PGx) <sup>18</sup> | | | < | | | | > | | | O | | 0 | | | | | | | | |

#Patients will record insulin usage for 7 days prior to out-patient visits (up to Month 24) and before telephone call/visit in Month 36 (if applicable) or final follow up.

Significant AEs including hypoglycaemic (≤3.9 mmol/L; ≤70 mg dL) and hyperglycaemic (>13.9 mmol/L; >250 mg/dL) events will be recorded in a diary whenever they occur, to include start and stop dates.

- 1. Patient admitted evening of Day -2
- 2. Discharged on Day 6 if health considered satisfactory by the investigator. Dosing Day 4-6 may be performed on out-patient basis


#### OTX116505

- 3. Physical exam performed to monitor for changes in clinical status
- 4. ECG pre-dose (in triplicate), at the end of the infusion and 6 hours post start infusion (if infusion < 6 hours)
- 5. Vital signs include temperature, blood pressure and pulse rate (in triplicate), and respiration rate
- 6. See Section 6.2.3 of the CSP for timings
- 7. Pre-dose on dosing days
- 8. If LFTs have shown an upward trend continue to monitor daily after day 6
- 9. HSV-1 & HSV-2 IgG & IgM will be measured at Day -1 and during the study if clinically indicated
- 10. If still positive at 6 months EBV viral load will be monitored every 3 months until month 24
- 11. One sample during visit
- 12. Blood samples for C-peptide and glucose levels collected at -10, 0, 15, 30, 60, 90 and 120 minutes
- 13. Plasma C-peptide and glucose levels will be measured during the hyperglycaemic clamp procedure at the following time points: L150, L165 and L180 minutes [during the euglycaemic (L)ow phase], H0, H60, H90, H120 and H140 minutes [during the hyperglycaemic (H)igh phase]
- 14. Mixed Meal and Glucose Clamp must be separated by at least 4 days
- 15. Patients will be asked to report verbally their HbA1c at Month 36 (if applicable) and/or final follow-up; followed eventually (if available) by a printed result via regular mail (or scan electronically).
- 16. Limited biomarkers on Day 6 pre-dose
- 17. Blood samples for exploratory biomarkers will only be analysed at Month 24 if indicated based on Month 12 results
- 18. One PGx (DNA) saliva sample taken between Day 1 and 6

# 11.1.4. Detail for Vitals, ECG and PK & PD Monitoring over the Infusion Period (Cohorts 1-4)

| Day | Cohort | Assessment | Pre<br>Dose | H 0 | 30 M | 1<br>H | 2 H | 3 H | 4 H | 5 H | Н 9 | 1 Н | Н 8 | Н 6 | 10 H | 11 H | 12 H | 13 H | 14 H | 15 H | 16 H |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Dosing | | | | | | | | | | | | | | | | | | | |
| | C1 | VItals <sup>1,2</sup> | X | X | | Х | Х | Х | X | Х | Х | X | X | Х | Х | X | X | Х | | | X |
| | 989,827 | ECG | X | | | | | | | | Х | | | X | | | | | | | |
| 2 | | PK/CD3 Saturation | Х | | Х | Х | Х | | Х | | Х | | Х | Х | | | | | | | Х |
| 1 | | Dosing | | | | | | | | | | | | | | | | | | | |
| | C2-C4 | Vitals <sup>1,2</sup> | X | X | | Х | Х | Х | Х | Х | Х | X | X | X | Х | X | Х | Х | Х | Х | Х |
| | | ECG | X | | | | | | | | Х | | | | | | Х | | | | |
| | | PK/CD3 Saturation | Х | | Х | Х | Х | | Х | | Х | | Х | | | | Х | | | | Х |
| | | Dosing | | | | | | | | | | | | | | | | | | | |
| | C1-C4 | Vitals <sup>1,2</sup> | X | X | | Х | Х | X | Х | Х | Х | X | X | Х | Х | | X | | | | Х |
| 2 | | ECG | X | | | | | | | | Х | | | | | | | | | | |
| | | PK/CD3 Saturation | Х | | | | | | | | | | | | | | | | | | |
| | | Dosing | | | | | | | | | | | | | | | | | | | |
| | C1-C4 | Vitals <sup>1,2</sup> | Х | Х | | Х | X | Х | Х | Х | Х | Х | Х | | | | Х | | | | X |
| 3 | 01101 | ECG | Х | | | | | Х | | | Х | | | | | | | | | | |
| | | PK/CD3 Saturation | Х | | | | | | | | | | | | | | | | | | |
#### OTX116505

| Day | Cohort | Assessment | Pre<br>Dose | Н 0 | 30 M | 1 H | 2 H | 3 H | 4 H | 5 H | Н 9 | 7 Н | 8 Н | Н 6 | 10 H | 11 H | 12 H | 13 H | 14 H | 15 H | 16 H |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 762 | | Dosing | | | | | 2536/4 | 7.00 | | 4/- | 25.44 | | | | 30 | | | | <b>V</b> = 0 | | |
| , | C1-C4 | Vitals <sup>1,2</sup> | X | X | | X | Х | X <sup>3</sup> | | | | | | | | | | | | | |
| 4 | | ECG | X | | | Х | | X <sup>3</sup> | | | | | | | | | | | | | |
| | | PK/CD3 Saturation | Х | | | | | | | | | | | | | | i | | | | |
| | | Dosing | | | | | | | | | | | | | | | | | | | |
| _ | C1-C4 | Vitals <sup>1,2</sup> | X | Х | | Х | Х | X <sup>3</sup> | | | | | | | | | | | | | |
| 5 | | ECG | Х | | | Х | | X <sup>3</sup> | | | | | | | | | | | | | |
| | | PK/CD3 Saturation | X | | | | | | | | | | | | | | | | | | |
| | | Dosing | | | | | | | | | | | | | | | | | | | |
| | | Vitals <sup>1,2</sup> | X | Х | | Х | Х | $X^3$ | , , | | | | | | | | | | | | |
| 6 | C1-C4 | ECG | X | | | Х | | X <sup>3</sup> | | | | | | | | | | | | | |
| | <u>L.</u> | PK/CD3 Saturation | X | | | Х | | | | | | | | | | | 4 | | | | |

- Blood pressure to be taken in triplicate at Pre-dose
   Vitals to be repeated at 30 min intervals should there be any safety concern
   If patients are dosed on an out-patient basis on Day 4, 5 and 6, vital signs and ECGs will stop after the 3 hour post dose time point (if the Investigator is satisfied with the clinical status of the patient), if there are any concerns then vital signs and ECGs may be continued as judged necessary by the investigator until the investigator is satisfied

| Day | Cohort | Assessment | Preferably within first hour of visit, time to be recorded in eCRF |
|---|---|---|---|
| 14 | C1-C4 | PK/CD3 Saturation | X |

# 11.2. Appendix 2: Assessment Windows

## 11.2.1. Definitions of Assessment Windows for Analyses

| Analysis Set / | Parameter | Target | Analysis | Window | Analysis<br>Timepoint |
|---|---|---|---|---|---|
| Domain | (if applicable) | | Beginning<br>Timepoint | Ending<br>Timepoint | |
| All | All | Nominal Day | Nominal<br>day – 1<br>days | Nominal<br>day + 1<br>days | Visits for<br>Day 14,<br>Day 21 and<br>Week 4<br>telephone<br>call |
| All | All | Nominal Day | Nominal day<br>-3 days | Nominal day<br>+3 days | Visits from<br>Week 6 to<br>Month 3 |
| All | All | Nominal Day | Nominal day<br>–7 days | Nominal day<br>+7 days | Visits from<br>Month 6 to<br>Month 24 |
| Safety/PK/CD 3 | All | In Window | -5 minutes predose | 0 minutes predose | Predose |
| Safety/PK/CD 3 | All | Nominal time point | Nominal time point | +5 minutes | Any<br>postdose up<br>to 6h |
| Safety/PK/CD 3 | All | Nominal time point | Nominal time point | +10 minutes | Any<br>postdose<br>after 6h |

Analysis Timepoint will be defined based on the nominal visit label, however a flag will be derived if a visit is considered outside of assessment window. Visits out of window will be included in all analyses but will be flagged in the listings. Sensitivity analyses may be performed excluding these visits.

# 11.3. Appendix 3: Study Phases

## 11.3.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to dosing.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Date of First Dose |
| During Dosing Date of First Dose <= Date <= Date of Final Dose + 1. | |
| Post-dose to Week 6 | Date of Final Dose + 1 < Date <= Date of Week 6 Visit <sup>[1]</sup> or Day 42 whichever is greater |
| Week 6 to Month 24 | Date of Week 6 Visit <sup>[1]</sup> or Day 42 whichever is greater < Date <= Month 24 visit. |
| Safety Follow-up | Date > Month 24 |
| [1] For participants who were consented Prior to Protocol Amendment 4, Day 42 will be used, as they will not have a Week 6 visit. | |

Note: for any rule that is relative to dose, the term date also includes time, if recorded. The end date for a visit as recorded in the SV domain will be used for the determining study phase.

#### 11.3.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and end date is prior to dosing |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Section 11.6 Premature Withdrawals & Handling of Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 11.4. Appendix 4: Data Display Standards & Handling Conventions

# 11.4.1. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Ratio to Baseline* | = Post-dose Visit Value / Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 5.2 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- \* only generated for strictly >0 parameters.

## 11.4.2. Reporting Process

| Re | porting Process | |
|---|---|---|
| So | ftware | |
| • | The currently supported versions of SAS will be used to perform all data analyses and generation of displays (tables, figures, and listings). | |
| Re | porting Area (GSK) | |
| > | HARP Server | UK1SALX00175 |
| > | HARP Area \\arwork\gsk2136525\otx116505\[reporting effort] \\arprod\gsk2136525\otx116505\[reporting effort] | |
| Re | porting Area (PXL) | |
| > | PXL Server | Kennet |
| A | SDTM Data | Transfer folder on Kennet |
| > | ADaM Data | Location: [project folder on kennet] /stats/nonversioncontrol/primary/data/sas/derived/main |
| > | The state of the s | |
| An | alysis Datasets | |
| AAA | > Define version 2.0 will be used for the SDTM datasets | |
| Ge | neration of RTF File | es |
| • | RTF files will be ge | nerated for the final reporting effort. |

#### 11.4.3. Reporting Standards

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.24: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Compiled Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables or figures.
- All unscheduled visits will be included in listings.

#### **Descriptive Summary Statistics**

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|------------------|--------------------------------------------|
| Categorical Data | N, n, frequency, % |

#### **Graphical Displays**

Refer to IDSL Compiled Statistical Principles 7.01 to 7.13.

#### 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

#### Multiple Measurements at One Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented, including the mean.
- The nominal time point will be used as described in Section 11.2.
- Participants having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date</li>
  - Ref Date ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### 11.5.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### Body Mass Index (BMI)

Calculated as Weight (kg) / [Height at screening (m)<sup>2</sup>

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula:
  - Duration of Exposure in Days = Treatment Stop Date (Treatment Start Date) + 1
- Participants who were randomized but did not report a treatment start date will be categorised
  as having zero days of exposure.
- The cumulative dose will be based on the formula:

### Cumulative Dose = Sum of doses on Day 1 to Day 6

- If there are any treatment breaks during the study, exposure data will be adjusted accordingly.
- In the calculation of daily infusion durations gaps between the two Day 1 syringes are included,
   i.e. duration will be calculated as end time of infusions start time of infusions.

#### 11.5.3. Safety

#### **ECG Parameters**

#### **RR** Interval

IF RR interval (msec) is not provided directly, then RR can be derived as:

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### Corrected QT Intervals

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### **Adverse Events**

#### General

| AE Type | Derivations |
|---|---|
| AE Onset Time<br>Since First Dose<br>(Days) | <ul> <li>If Treatment Start Date &gt; AE Onset Date : = AE Onset Date - Treatment Start Date</li> <li>If Treatment Start Date ≤ AE Onset Date : = AE Onset Date - Treatment Start Date + 1</li> <li>Missing otherwise</li> </ul> |
| AE Duration (Days) | > AE Resolution Date - AE Onset Date + 1 |
| AE = Drug-related | If relationship is marked 'YES' on eCRF OR value is missing. |

### Adverse Events: CRS and Clinical Symptoms of Mononucleosis Definition

- The current MedDRA version at time of database lock will be used for coding of AE's.
- AEs considered to be related to CRS during the first 14 days post first dose will be determined by medical expert review conducted by the GSK team.
- For reporting of clinical symptoms of mononucleosis, the following AE's will be extracted based on Preferred Term. In addition, other terms maybe included at the time of reporting.

| Reporting | Preferred Term | Verbatim Terms |
|-----------|----------------|----------------------------|
| Clinical | Fatigue | Feeling tired & Low energy |

| Adverse Events | | |
|---|---|---|
| General | | |
| Symptoms of | Malaise | Feeling unwell |
| Mononucleosis | Myalgia | Joint and muscle pain & Flu like symptoms |
| | Oropharyngeal pain | Sore throat, throat pain |
| | Lymphadenopathy | Swollen glands |
| | Pyrexia | High temperature, Feeling hot and cold & Shivering |

## **Laboratory Parameters**

- All BLQ values will be imputed with ½ LLOQ.
- All ALQ values will be imputed with the ALQ + [smallest positive number with the same number
  of decimal places as the ALQ is reported with]
- Values reported as < x are assumed to have an LLOQ of x.</li>
- Values reported as > x are assumed to have an ALQ of x.

#### **EBV**

- EBV Serology:
  - Categories (negative, positive) will be derived from absolute IgG and IgM values according to a worst case approach from absolute virus results

| | QUEST Classification of INDEX | Quest<br>classification of<br>U/ml | BDR Classification of AE/mL | Unified Classification |
|---|---|---|---|---|
| IgG | < OR = 0.90 NEGATIVE<br>0.91 - 1.09 EQUIVOCAL<br>> OR = 1.10 POSITIVE | | negative : <20 positive : 20 or more | NEGATIVE<br>POSITIVE<br>POSITIVE |
| IgM | < OR = 0.90 NEGATIVE | negative: <36 | negative : <20<br>weakly positive : 20-40 | NEGATIVE<br>POSITIVE |
| | 0.91 - 1.09 EQUIVOCAL<br>> OR = 1.10 POSITIVE | positive: 36 or more | positive : 40 or more | POSITIVE<br>POSITIVE |

- EBV Viral Load (EBVPCR\_B):
  - Viral Load will also be categorized, using these groups:
    - 0-1000 copies/10^6PBM cells
    - >1000-10000 copies/10^6PBM cells
    - >10000-100000 copies/10^6PBM cells
    - >100000 copies/10^6PBM cells
  - The sames rules as for laboratory parameters will be applied for BLQ/ALQ values.

Any viral load given as > XX.X or < XX.X will be treated in the same manner as described for laboratory parameters. If the result is given as not detected, then it will be imputed as 1 copies/10^6PBM cells instead.

#### **Auto-Antibodies**

Positive/Negative results will be derived for all the auto-antibodies, where positive is defined as:

- antibody to glutamic acid decarboxylase (anti-GAD) ≥ 2.6% binding
- antibody to protein tyrosine phosphatase-like protein (anti IA 2) ≥ 0.44% binding
- Qualitative status (positive/negative status) is directly provided for islet cell antigen and will be used
- ZnT8 Autoantibody ≥ 1.02% binding
- IAA ≥ 0.6% binding

In addition, the number of positive results at Screening (with the exception of IAA) will be derived in ADSL.

### **Immunogenicity**


OTX116505

The presence of anti-drug antibodies will be summarized by positive/negative status at each time point. A participant is considered positive at a specific time point if both the Screening and the Confirming sample is positive.

The listing will show individual results for the Screening, Confirming and Titer tests. Not applicable tests will be omitted from the listing.

### 11.5.4. Efficacy

#### Weighted Means AUC (MMTT & Hyperglycemic Clamp Test)

The weighted mean parameters will be derived by calculating the area under the curve (AUC) using the trapezoidal rule, and then dividing by the actual relevant time interval (i.e. t<sub>f</sub> - t<sub>i</sub>):

Weighted Mean (t<sub>f</sub>-t<sub>i</sub>) = 
$$\left[\frac{1}{2}\sum_{i=1}^{I-1}(t_{i+1}-t_i)(y_i+y_{i+1})\right]/[tl-tf]$$

Where (example provided for MMTT AUC(0-120m):

- $y_i$  = Value of endpoint at i<sup>th</sup> time point
- $t_i$  = The i<sup>th</sup> actual time point (mins) for MMTT:
  - Before MMTT: t<sub>1</sub>=0
  - After MMTT : t<sub>2</sub> =15m, t<sub>3</sub> = 30m, t<sub>4</sub>=60m, t<sub>5</sub>=90m, t<sub>6</sub>=120m
- tf = Actual time point (hrs) of first non-missing obs (e.g. in planned time tf=0h)
- tl = Actual time point (hrs) of last non-missing obs (e.g. in planned time tl=120m)
- I = Number of time points used in the AUC calculation (e.g. I=6)
- The examples provide details of how AUC's are calculated under certain scenario's and is to be adapted based on the study endpoints:



# Weighted Means AUC (MMTT & Hyperglycemic Clamp Test)

| Profile | Weighted Mean AUC Derivation |
|---|---|
| Complete | Area / Complete Time Interval |
| First Time Point Missing | Remaining Area / Remaining Time Interval |
| Last Time Point Missing | Remaining Area / Remaining Time interval |
| Time Point Missing Within Profile | Area using values of Remaining Profile / Complete Time Interval |

#### Efficacy

#### Hyperglycemic Clamp Test: Calculation of Insulin Sensitivity Index (ISI)

The ISI during the hyperglycemic phase (120-140 min) of the hyperglycemic clamp test (HCT) (Defronzo et al, 1979) will be calculated as:

$$ISI = (M / I)_{120-140min} \times 100 (a)$$

- ➤ Ratio of glucose metabolized between 120 & 140 min (M expressed as mmol.kg-1.min-1) **AND** average insulin concentration between 120 & 140 min (I expressed as pmol/I), multiplied by 100.
- As the average insulin concentration is not directly available in the data, it will be replaced with the average C-peptide concentration instead.
- The glucose values taken for the derivation are those measured in the laboratory samples (LBSCAT = CLAMP), not the bedside glucose values (LBSCAT = BEDSIDE GLUCOSE).
- ➤ To correct for minor blood glucose fluctuations, M will be calculated as the average glucose infusion rate between 120 and 140 min minus a "space correction".
- Parameter M & I will be derived as follows:

#### Parameter = M

$$M = INF - SC(b)$$

- ➤ M = Amount of glucose metabolized during the last 20 minutes (120-140 min) of the hyperglycemic phase of the HG clamp test.
- ➤ M expressed as mmol.kg-1.min-1.
- ➤ INF: Glucose infusion rate (mmol.kg<sup>-1</sup>.min<sup>-1</sup>).
- > SC: Glucose space correction, amount of glucose necessary to fill the plasma glucose equivalent space (mg.kg-1.min-1):

$$SC = (G2 - G1) \times 0.095 (c)$$

- ✓ G2 and G1 are the glucose concentrations in milligrams per deciliter at the end and at the beginning of the time period.
- ✓ The value for **SC** needs to be converted to mmol.kg<sup>-1</sup>.min<sup>-1</sup> before filling in (b).

#### Parameter = I

Average C-peptide concentration during the same period (120-140 min) (expressed as pmol/l).

#### NOTES:

- [1] Following review of the data for missing values, ISI may be calculated using the average C-peptide concentrations instead of average insulin concentrations between 120-140 min.
- [2] Following review of the data, HOMA-2IR during HCT at following time points: -180 min (L180), -165 min (L165) and -150 min (L150) and during MMTT at time points: -10 min and 0 min (Matthews et al, 1985; Levy et al, 1998) may be also be calculated.

#### Efficacy

#### Mean Daily Insulin Use

- The mean daily insulin use in IU/kg will be derived as follow:
  - Sum doses by participant and day to get daily dose in IU
  - 2. Missing daily doses during the seven day space will be imputed with 0
  - Take the average and divide by the most recent available weight measurement to get mean daily insulin use in IU/kg

#### Responders (HbA1c)

- A participant will be considered a responder if, at a given visit, the participant has:
  - HbA1c ≤7.0% and
  - Mean daily insulin use < 0.5 units/kg/day.</li>
- HbA1c and mean daily insulin use will be calculated as described above, and values compared
  at each time point of interest (Week 4, 8, 16, 28, 40, 52 and 64) to determine if a participant is
  classed as a responder or not

#### **Partial Remission Status**

- A participant achieving partial remission status is defined as a participant with Insulin Dose Adjusted A1c (IDAA1C) ≤9.0 [3]
- Insulin-dose adjusted A1c (IDAA1c) is a composite variable, which is a weighted sum of insulin
  use and HbA1c level.
- IDAA1C is calculated as:
  - HbA1c(%) + 4 x{mean daily insulin use per kg body weight (IU/kg)}
  - where the computation of mean total daily insulin use per kg body weight is as described above
- The calculated IDAA1C value will be rounded to 2 decimal places before assigning partial remission status. Therefore the largest value assigned as ≤9.0 would be 9.004999.

### C-peptide Responder

- A participant is considered a C-peptide responder if there is > -40% change from baseline in C-peptide MMTT Weighted Mean AUC at 24 months (so participants with >40% loss in C-peptide are non-responders) [10]
- Participants with missing C-peptide values at 24 months or baseline will have a missing C-peptide responder state. They will be reported as such in frequency tabulations, but not included in figures by C-peptide responder status.

•

# 11.5.5. Pharmacodynamics

# **Target Engagement**

## Overview of CD3 SAT/MOD Target Engagement Parameters

The following parameters will be listed only:

| Parameter Category 1 | LBTESTCD | LBTEST |
|----------------------|----------|---------------------------------|
| CD3 SAT/MOD | CD4 | CD4 |
| CD3 SAT/MOD | CD4LY | CD4/Lymphocytes |
| CD3 SAT/MOD | CD8 | CD8 |
| CD3 SAT/MOD | CD8LY | CD8/Lymphocytes |
| CD3 SAT/MOD | MLYMP | Acquired Lymphocyte Events Mean |
| CD3 SAT/MOD | CD3EFS1 | CD3e Free MESF(CD4+) |
| CD3 SAT/MOD | CD3EFS2 | CD3e Free MESF(CD8+) |
| CD3 SAT/MOD | CD3EBS1 | CD3e Bound MESF(CD4+) |
| CD3 SAT/MOD | CD3EBS2 | CD3e Bound MESF(CD8+) |

The following parameters will be summarised:

| CD3 SAT/MOD | CD3ER8 | CD3e Copies/Cell(CD4+) |
|-------------|---------|------------------------------|
| CD3 SAT/MOD | CD3ER9 | CD3e Copies/Cell(CD8+) |
| CD3 SAT/MOD | CD3EFR8 | CD3e Free Copies/Cell(CD4+) |
| CD3 SAT/MOD | CD3EFR9 | CD3e Free Copies/Cell(CD8+) |
| CD3 SAT/MOD | CD3EBR8 | CD3e Bound Copies/Cell(CD4+) |
| CD3 SAT/MOD | CD3EBR9 | CD3e Bound Copies/Cell(CD8+) |

#### Calculation of Target Engagement (%)

The following formulas will be used to derive the Target Engagement percentage:

Total Binding Sites = Occupied Binding Sites + Free Binding Sites + Down Modulated Binding Sites

In this equation, Total Binding Sites is not equal to the corresponding parameter shown above (e.g. CD3ER8 for CD4), except for the Baseline Visit. Instead, they differ by the number of Down Modulated Binding Sites, which is presumed to be zero at Baseline.

As the Total Binding Sites can be assumed to be approximately constant, the number of Down Modulated Binding Sites can be derived as follows:

Down Modulated Binding Sites at Visit X

= Total Binding Sites at Baseline - Total Binding Sites at Visit X

Therefore, percentage Target Engagement can be estimates as follows:

$$\text{Target Engagement (\%)} = \frac{\text{Occupied Binding Sites Visit X} + \text{Down Modulated Binding Sites Visit X}}{\text{Total Binding Sites at Baseline}} \times 100$$

Target Engagement will be derived using 'Copies/Cell'for both CD4 and CD8, but not for MESF values, as the corresponding values have not been measured consistently across cohorts.

#### **Derived Target Engagement (%) Parameters**

| | arameter<br>ategory 1 | Parameter<br>Code | Parameter |
|---|---|---|---|
| CD3 S | SAT/MOD | CD4TE | Otelixizumab Down Modulation and Receptor Occupancy of CD3 ^{unicode epsilon} Target Sites on CD4 |
| CD3 S | SAT/MOD | CD8TE | Otelixizumab Down Modulation and Receptor Occupancy of CD3 ^{unicode epsilon} Target Sites on CD8 |

# 11.6. Appendix 6: Premature Withdrawals & Handling of Missing Data

#### 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>As defined in the protocol the overall study duration for each participant is 36 months (up to 36 months including the screening period).</li> </ul> |
| | <ul> <li>Primary study completion for each participant will be at 24 months when all<br/>available data will be analysed.</li> </ul> |
| | <ul> <li>Participant study completion is defined as participants who either prematurely<br/>withdrawn or:</li> </ul> |
| | <ul> <li>Patients who had yet to complete their Month 24 visit at the time of<br/>approval of Protocol Amendment 9, will be defined as completed if they<br/>complete the Month 24 Visit.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>Patients past Month 24 visit at time of approval of Protocol Amendment 9 will<br/>be followed up with a final communication or visit (final follow up) and will be<br/>defined as completors if they have completed this follow-up visit. Withdrawn<br/>participants maybe replaced in the study.</li> </ul> |
| | <ul> <li>All available data from participants who were withdrawn from the study will be<br/>listed and all available planned data will be included in summary tables and<br/>figures, unless otherwise specified. If data is present after the participants<br/>withdrawal from treatment date, this data will be flagged in the listings.</li> </ul> |

# 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | <ul> <li>Any participants excluded from the summaries and/or statistical analyses will be<br/>documented along with the reason for exclusion in the clinical study report.</li> </ul> |

# 11.6.3. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 11.7. Appendix 7: Values of Potential Clinical Importance

# 11.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Basophiles | x109/ L | | 0.02 | 0.1 |
| Hamataarit | Datis of 1 | | 0.24 | 0.54 |
| Hematocrit | Ratio of 1 | Δ from BL | ↓0.075 | |
| Haman makin | a.7a11 | | 8 | 18 |
| Hemoglobin | g/dL | Δ from BL | ↓2.5 | |
| Lymphocytes | x109/ L | | 0.8 | |
| Mean Corpuscular Volume (MCV) | fL | | 80 | 100 |
| Mean Corpuscular Hemoglobin (MCH) | pg | | 27 | 33 |
| Mean Corpuscular Hemoglobin Concentration (MCHC) | g/L | | 330 | 360 |
| Monocytes | x109/L | | 0.2 | 1.0 |
| Eosinophils | x109/L | | | 0.44 |
| Neutrophil Count | x109/L | | 1.5 | |
| Platelet Count | x109/L | | 100 | 550 |
| Red Blood Cell Count (RBC) | x10 <sup>12</sup> /L | | 4.2 | 5.9 |
| Reticulocyte Count | x109/L | | 23 | 90 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | 3/8 3/9/2 |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | | | 1.3x ULN |
| | | $\Delta$ from BL | | ↑ 44 |
| Glucose | mmol/L | | 3 | 11.1 |
| Potassium | mmol/L | | 3.2 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |

| Liver Function | | | |
|----------------|-------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |

| Liver Function Test Analyte | Units | Catogory | Clinical Concern Range |
|---|---|---|---|
| Test Analyte | Units | Category | |
| ALT/SGPT | IU/L | High | ≥ 2x ULN |
| | | | ≥ 3x ULN |
| AST/SGOT | IU/L | High | ≥ 2x ULN |
| Alkaline Phosphatase | IU/L | High - | ≥ 1.5x ULN |
| Alkaline i nospilatase | IO/L | Tilgit | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | ≥ 1.5xULN T. Bilirubin + ≥ 2x ULN ALT |
| T. Bilirubin + ALT | | High | |
| | U/L | 100 | $\geq$ 2xULN T. Bilirubin + $\geq$ 3x ULN ALT |
| Urea Nitrogen (BUN) | | Low | < 2.9 |
| | mmol/L | High | >7.1 |
| | | Low | < 98 |
| Chloride | mmol/L | High | |
| | , 100 | High | ≥ 2x ULN |
| Direct Bilirubin | μmol/L | High | > 7.1 |
| Urata | umo!/l | Low | < 150 |
| Urate | μmol/L | High | > 470 |
| Total Protein | g/l | Low | < 60 |
| TUIAI FTUICIII | g/L | High | > 78 |

# 11.7.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | * * | 100 (100 m) (100 m) | elle State S |
| Absolute QTc Interval | msec | | >450 |
| Absolute PR Interval | msec | < 110 | > 220 |
| Absolute QRS Interval | msec | < 75 | > 120 |
| Change from Baseline | -0 19 | | |
| Increase from Baseline QTc | msec | >60 | |

# 11.7.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |
| Respiration Rate | Min-1 | < 10 | > 30 |

# 11.8. Appendix 8: Biomarker Analyses

## 11.8.1. Handling of duplicate data due to reruns

Due to a rerun of samples from cohorts 1 and 2, duplicate data may be included in the SDTM data. For any such case, only the newer data will be used for summaries and the older data will only be included (with flag) in the listings.

# 11.8.2. Frequency and phenotype of lymphocyte subsets by flow cytometry

The list of analytes below will be summarised and analysed as per Section 9.4

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Der<br>ive<br>d | Details |
|---|---|---|---|---|
| Lymphocytes | LYM | 10^9 /L | u | |
| CD3 | CD3 | 10^9 /L | | CD3 T cells (10^9/L) |
| CD3/Lymphocytes | CD3LY | % | | CD3 T cells |
| CD4 | CD4 | 10^6 /L | | CD4 T cells (10^6/L) |
| CD4/Lymphocytes | CD4LY | % | | CD4 T cells |
| CD8 | CD8 | 10^6 /L | | CD8 T cells (10^6/L) |
| CD8/Lymphocytes | CD8LY | % | | CD8 T cells |
| CD19 | CD19 | 10^9 /L | | B cells (10^9/L) |
| CD19/Lymphocytes | CD19LY | % | | B cells |
| CD4+CXCR3+CCR6-/CD4+ | CDX5554 | % | | Th1 |
| CD4+CXCR3+CCR6- | CDX555C | 10^6 /L | Yes | [CDX5554] x [CD4] / 100 |
| CD4+CXCR3-CCR6-/CD4+ | CDX5564 | % | | Th2 |
| CD4+CXCR3-CCR6- | CDX556C | 10^6 /L | Yes | [CDX5564] x [CD4] / 100 |
| CD4+CXCR3-CCR6+/CD4+ | CDX5574 | % | | Th17 |
| CD4+CXCR3-CCR6+ | CDX557C | 10^6 /L | Yes | [CDX5574] x [CD4] / 100 |
| CD4+CXCR3+CCR6+/CD4+ | CDX5584 | % | | Th1 andTh17 |
| CD4+CXCR3+CCR6+ | CDX558C | 10^6 /L | Yes | [CDX5584] x [CD4] / 100 |
| CD4+CD25+CD127-/CD4+ | CDX5594 | % | | CD4 Tregs |
| CD4+CD25+CD127- | CDX559C | 10^6 /L | Yes | [CDX5594] x [CD4] / 100 |
| CD8+CXCR3+CCR6-/CD8+ | CDX5618 | % | | Tc1 |
| CD8+CXCR3+CCR6- | CDX561C | 10^6 /L | Yes | [CDX5618] x [CD8] / 100 |
| CD8+CXCR3-CCR6-/CD8+ | CDX5628 | % | | Tc2 |
| CD8+CXCR3-CCR6- | CDX562C | 10^6 /L | Yes | [CDX5628] x [CD8] / 100 |
| CD8+CXCR3-CCR6+/CD8+ | CDX5638 | % | | Tc17 |
| CD8+CXCR3-CCR6+ | CDX563C | 10^6 /L | Yes | [CDX5638] x [CD8]) / 100 |
| CD8+CXCR3+CCR6+/CD8+ | CDX5648 | % | | Tc1/ Tc17 |
| CD8+CXCR3+CCR6+ | CDX564C | 10^6 /L | Yes | [CDX5648] x [CD8] / 100 |
| CD8+CD25+CD127-/CD8+ | CDX5668 | % | | CD8 Tregs |
| CD8+CD25+CD127- | CDX566C | 10 ^6/L | Yes | [CDX5668] x [CD8] / 100 |
| CD8+CD45RA-/CD8+ | CDX5118 | % | | CD8 Memory |
| CD8+CD45RA+/CD8+ | CDX1688 | % | | CD8 Naive |
| CD8-CD45RA-/CD8- | CDX601C8 | % | | CD4 Memory |
| CD8-CD45RA+/CD8- | CDX602C8 | % | | CD4 naïve |

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Der<br>ive<br>d | Details |
|---|---|---|---|---|
| CD8 Memory<br>Exhausted(CD45RA-CD8+) | CDX569J9 | % | | CD3+CD8+CD45RA-EOMES+ TIGIT+<br>KLRG1+ (% of CD45RA-CD8+) |
| CD8 Mem Exhausted IL-<br>6R/CD8 Mem Exhaustd | CDX570K1 | % | | CD3+CD8+CD45RA-EOMES+ TIGIT+<br>KLRG1+ CD126+ (% of<br>CD3+CD8+CD45RA-EOMES+ TIGIT+<br>KLRG1+) |
| CD8 Mem Exhausted IL-6R<br>MNFI of CD126 | CDX570J8 | count | | CD3+CD8+CD45RA-EOMES+ TIGIT+<br>KLRG1+ CD126+ (CD126 MFI) |
| CD3+CD8+CD126+/CD8+ | CDX5678 | % | | CD8 IL-6R |
| CD3+CD8+CD126+ MNFI of CD126 | CDX567J8 | count | | CD8 IL-6R |
| CD3+CD8-CD126+/CD8- | CDX568C8 | % | 1 | CD4 IL-6R |
| CD3+CD8-CD126+ MNFI of CD126 | CDX568J8 | count | | CD4 IL-6R |
| CD3+CD8+CD45RA+CD12<br>6+ MNFI of CD126 | CDX571J8 | count | | CD8 naive IL-6R |
| CD3+CD8+CD45RA-<br>CD126+ MNFI of CD126 | CDX572J8 | count | | CD8 memory IL-6R |
| CD3+CD8-<br>CD45RA+CD126+ MNFI of<br>CD126 | CDX573J8 | count | | CD4 naive IL-6R |
| CD3+CD8-CD45RA-<br>CD126+ MNFI of CD126 | CDX574J8 | count | | CD4 memory IL-6R |

For ADLB PARAMCD will be set to be the same as LBTESTCD and PARAM will be set to LBTEST concatenated with the unit in brackets (in case of counts, no unit will be added).

# 11.8.3. Percentage of CD3 cells, FoxP3 regulatory cells and TH17 cells by epigenetic quantification

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Unit | Deri<br>ved | Details |
|---|---|---|---|---|
| CD3+/Total Cells | CD3CE | % | | |
| FoxP3/Total Cells | FOXP3CE | % | | |
| T Helper 17 Cells/Total Cells | TH17CE | % | | |
| FoxP3/CD3+ | FOXP3CD3 | % | Yes | = [FOXP3CE] x 100/[CD3CE] |
| T Helper 17 Cells/CD3+ | TH17CD3 | % | Yes | = [TH17CE] x 100/[CD3CE] |

# 11.8.4. Frequency and phenotype of HLA-A2-resticted antigen-specific CD8+ T cells by multimer analysis

The data for the Frequency and phenotype of HLA-A2-resticted antigen-specific CD8+ T cells by multimer analysis will be reported only for the HLA-A2 Positive population.

Visits where the CD8 count is less 30,000 cells will be excluded from analysis and listed only except for EBV-specific CD8+ T cells for which counts less than 15,000 will be excluded from analysis and listed only. CD8 counts between 30,000 – 50,000 cells will be included in summaries but flagged in listings. Parameters will only be summarised if >40% of baseline visits and >40% of post-baseline visits are evaluable for that parameter.

The list of analytes below are for classification of participants and for determining the quality of cells, and hence will be listed only.

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Deri<br>ved | Details |
|---|---|---|---|---|
| Viable Cells Count | VIABCC | Count | | |
| Viable Cells/Total Cells | VIABCCE | % | | |
| CD8+ Count | CD8C | Count | | |

The list of analytes below will be summarised and analysed as per Section 9.1.1.2.

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Deri<br>ved | Details |
|---|---|---|---|---|
| T1D-specific CD8 T<br>Cells/CD8+ | T1D8CD8 | % | | |
| T1D-specific CD8 T Cells | T1DCD8 | 10^6/L | Yes | [T1D8CD8]*[CD8] / 100 |
| Insulin B10-18-specific CD8<br>T Cells/CD8+ | B1018C88 | % | | |
| Insulin B10-18-specific CD8<br>T Cells | B1018C8 | 10^6/L | Yes | [B1018C88] * [CD8] / 100 |
| PPI-specific CD8 T<br>Cells/CD8+ | PPICD88 | % | | |
| PPI-specific CD8 T Cells | PPICD8 | 10^6/L | Yes | [PPICD88] * [CD8] / 100 |
| Novel Insulin Epitope CD8 T<br>Cells/CD8+ | NINECD88 | % | | |
| Novel Insulin Epitope CD8 T<br>Cells | NINECD8 | 10^6/L | Yes | [NINECD88] * [CD8] / 100 |
| GAD65-specific CD8 T<br>Cells/CD8+ | GD65CD88 | % | | |
| GAD65-specific CD8 T Cells | GD65CD8 | 10^6/L | Yes | [GD65CD88] * [CD8] / 100 |
| IGRP-specific CD8 T<br>Cells/CD8+ | IGRPCD88 | % | | |
| IGRP-specific CD8 T Cells | IGRPCD8 | 10^6/L | Yes | [IGRPCD88] * [CD8] / 100 |
| IA2-specific CD8 T<br>Cells/CD8+ | IA2CD88 | % | | |
| IA2-specific CD8 T Cells | IA2CD8 | 10^6/L | Yes | [IA2CD88] * [CD8] / 100 |

| Lab Test | Lab Test | Units | Deri | Details |
|---|---|---|---|---|
| (LBTEST) | (LBTESTCD) | | ved | |
| ppIAPP-specific CD8 T<br>Cells/CD8+ | PIAPCD88 | % | | |
| ppIAPP-specific CD8 T Cells | PIAPCD8 | 10^6/L | Yes | [PIAPCD88] * [CD8] / 100 |
| ZnT8-specific CD8 T | ZNT8CD88 | % | 100 | [1111 0200] [020]7 100 |
| Cells/CD8+ | | | | |
| ZnT8-specific CD8 T Cells | ZNT8CD8 | 10^6/L | Yes | [ZNT8CD88] * [CD8] / 100 |
| A2-specific CD8 T<br>Cells/CD8+ | A2CD8CD8 | % | | |
| A2-specific CD8 T Cells | A2CD8 | 10^6/L | Yes | [A2CD8CD8] * [CD8] / 100 |
| EBV-specific CD8 T<br>Cells/CD8+ | EBVCD88 | % | | |
| EBV-specific CD8 T Cells | EBVCD8 | 10^6/L | Yes | [EBVCD88] * [CD8] / 100 |
| CXCR3+ T1D-specific CD8 T<br>Cells/CD8+ | CDX5388 | % | | Migratory T1D-specific cells/ total CD8 cells |
| CXCR3+ T1D-specific CD8 T<br>Cells | CDX538C | 10^6/L | Yes | [CDX5388] * [CD8] / 100 |
| CCR7+CD45RA+ T1D CD8+ | CDX543J6 | % | | Naive T1D-specific cells / total T1D- |
| Cells/T1D CD8 | ODV5 400 | 4040// | 1 1/ | specific cells |
| CCR7+CD45RA+ T1D CD8<br>T Cells | CDX543C | 10^6/L | Yes | [CDX543J6] * [T1DCD8] / 100 |
| CCR7+CD45RA- T1D CD8+<br>Cells/T1D CD8 | CDX544J6 | % | | Central memory T1D-specific cells / total T1D-specific cells |
| CCR7+CD45RA- T1D CD8 T<br>Cells | CDX544C | 10^6/L | Yes | [CDX544J6] * [T1DCD8] / 100 |
| CCR7-CD45RA- T1D CD8+<br>Cells/T1D CD8 | CDX545J6 | % | | Effector T1D-specific cells / total T1D-<br>specific cells |
| CCR7-CD45RA- T1D CD8+<br>T Cells | CDX545C | 10^6/L | Yes | [CDX545J6] * [T1DCD8] / 100 |
| CCR7-CD45RA+ T1D CD8+<br>Cells/T1D CD8 | CDX546J6 | % | | Terminally differentiated effector memory T1D-specific cells / total T1D-specific cells |
| CCR7-CD45RA+ T1D CD8 T | CDX546C | 10^6/L | Yes | [CDX546J6] * [T1DCD8] / 100 |
| Cells | 02/10/100 | 10 0/2 | 100 | [ebxercool [ribebel/ite |
| CCR7+CD45RA+CXCR3+T1<br>D CD8 T Cell/T1D CD8 | CDX539J6 | % | | Migratory Naive T1D-specific cells / total T1D-specific cells |
| CCR7+ CD45RA+<br>CXCR3+T1D CD8 T Cell | CDX539C | 10^6/L | Yes | [CDX539J6] * [T1DCD8] / 100 |
| CCR7+CD45RA-CXCR3+<br>T1D CD8+ Cell/T1D CD8 | CDX540J6 | % | | Migratory Central memory T1D-specific cells / total T1D-specific cells |
| CCR7+CD45RA-CXCR3+ | CDX540C | 10^6/L | Yes | [CDX540J6] * [T1DCD8] / 100 |
| T1D CD8 T Cells | ODVE4410 | 0/ | | Missatas Effects TAD 25 25 21 11 11 |
| CCR7-CD45RA-CXCR3+<br>T1D CD8+ Cell/T1D CD8 | CDX541J6 | % | | Migratory Effector T1D-specific cells / total T1D-specific cells |
| CCR7-CD45RA-CXCR3+<br>T1D CD8 T Cells | CDX541C | 10^6/L | Yes | [CDX541J6] * [T1DCD8] / 100 |
| CCR7-CD45RA+CXCR3+<br>T1D CD8+ Cell/T1D CD8 | CDX542J6 | % | | Migratory Terminally differentiated effector memory T1D-specific cells / total T1D-specific cells |
| CCR7-CD45RA+CXCR3+ | CDX542C | 10^6/L | Yes | [CDX542J6] * [T1DCD8] / 100 |

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Deri<br>ved | Details |
|---|---|---|---|---|
| T1D CD8 T Cells | | | | |
| CCR7+CD45RA+ EBV CD8+<br>Cells/EBV CD8 | CDX551J7 | % | | Naive EBV -specific cells / total EBV-<br>specific cells |
| CCR7+CD45RA+ EBV CD8<br>T Cells | CDX551C | 10^6/L | Yes | [CDX551J7] * [EBVCD8] / 100 |
| CCR7+CD45RA- EBV CD8+<br>Cells/EBV CD8 | CDX552J7 | % | | Central memory EBV-specific cells / total EBV-specific cells |
| CCR7+CD45RA- EBV CD8 T<br>Cells | CDX552C | 10^6/L | Yes | [CDX552J7] * [EBVCD8] / 100 |
| CCR7-CD45RA-EBV CD8+<br>Cells/EBV CD8 | CDX553J7 | % | | Effector EBV-specific cells / total EBV-specific cells |
| CCR7-CD45RA-EBV CD8 T<br>Cells | CDX553C | 10^6/L | Yes | [CDX553J7] * [EBVCD8] / 100 |
| CCR7-CD45RA+ EBV CD8+<br>Cells/EBV CD8 | CDX554J7 | % | | Terminally differentiated effector memory EBV-specific cells / total EBV-specific cells |
| CCR7-CD45RA+ EBV CD8 T<br>Cells | CDX554C | 10^6/L | Yes | [CDX554J7] * [EBVCD8] / 100 |
| CCR7+CD45RA+CXCR3+<br>EBV CD8+ Cell/EBV CD8 | CDX546J7 | % | | Migratory Naive EBV-specific cells / total EBV-specific cells |
| CCR7+CD45RA+CXCR3+<br>EBV CD8 T Cells | CDX547C | 10^6/L | Yes | [CDX546J7] * [EBVCD8] / 100 |
| CCR7+CD45RA-CXCR3+<br>EBV CD8+ Cell/EBV CD8 | CDX548J7 | % | | Migratory Central memory EBV-specific cells / total EBV-specific cells |
| CCR7+CD45RA-CXCR3+<br>EBV CD8 T Cells | CDX548C | 10^6/L | Yes | [CDX548J7] * [EBVCD8] / 100 |
| CCR7-CD45RA-CXCR3+<br>EBV CD8+ Cell/EBV CD8 | CDX549J7 | % | | Migratory Effector EBV-specific cells / total EBV-specific cells |
| CCR7-CD45RA-<br>CXCR3+EBV CD8 T Cell | CDX549C | 10^6/L | Yes | [CDX549J7] * [EBVCD8] / 100 |
| CCR7-CD45RA+CXCR3+<br>EBV CD8+ Cell/EBV CD8 | CDX550J7 | % | | Migratory Terminally differentiated effector memory EBV-specific cells / total EBV-specific cells |
| CCR7-CD45RA+CXCR3+<br>EBV CD8 T Cells | CDX550C | 10^6/L | Yes | [CDX550J7] * [EBVCD8] / 100 |

# 11.8.5. Frequency of interferon-gamma- secreting antigen-reactive cells by ELISPOT

The list of analytes below are for classification of participants and for determining the quality of cells, and hence will be listed only.

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Derived | Details |
|---|---|---|---|---|
| Viable Cells Count | VIABCC | Count | | |
| Viable Cells/Total Cells | VIABCCE | % | | |

The list of analytes below will listed. PARAM/PARAMCD will be created from LBTEST/LBTESTCD and the stimulus (e.g. EBV) which is stored in SUPPLB.

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Derived | Details |
|---|---|---|---|---|
| Interferon Gamma Spot<br>Forming Cell Count | IFNGSFCC | count/10 <sup>^</sup><br>6PBMC | | |

The following stimulants have been used:

- Unstimulated
- GAD Glutamic Acid Decarboxylase
- icIA-2 Intracellular Islet Antigen-2
- EBV Epstein Barr Virus
- PI Pro-insulin
- PI C-pep Pro-insulin-derived C-peptide
- PPI Leader Prepro-insulin Leader

# 11.8.6. Quantification of serum cytokines and soluble cytokine receptors

The list of analytes below will be summarised and analysed as per Section 9.4.

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Derived | Details |
|---|---|---|---|---|
| Interferon Gamma (ng/L) | IFNG | (ng/L) | | |
| Soluble Interleukin<br>6 Receptor<br>(ng/mL) | IL6SR | (ng/mL) | | |
| Interleukin 6<br>Signal Transducer<br>(ng/mL) | IL6ST | (ng/mL) | | Soluble gp130 |
| Interleukin 10<br>(ng/L) | INTLK10 | (ng/L) | | |
| Interleukin 12<br>(ng/L) | INTLK12 | (ng/L) | | |
| Interleukin 13<br>(ng/L) | INTLK13 | (ng/L) | | |
| Interleukin 1 Beta (ng/L) | INTLK1B | (ng/L) | | |
| Interleukin 2 (ng/L) | INTLK2 | (ng/L) | | |
| Interleukin 4 (ng/L) | INTLK4 | (ng/L) | | |
| Interleukin 6 (ng/L) | INTLK6 | (ng/L) | | |
| Interleukin 8 (ng/L) | INTLK8 | (ng/L) | | |

## 11.8.7. TCR deep sequencing

The list of analytes below will be summarised and analysed as per Section 9.1.1.2.

| Test (PFTEST) | Test Code<br>(PFTESTCD) | Units | Derived | Details |
|----------------------|-------------------------|-------|---------|---------|
| Productive Clonality | AH001 | % | Ì | |

Further TCR deep sequencing endpoint may be explored through Adaptive Biotechnology's ImmunoSeq<sup>TM</sup> Analyser but these are considered as further exploratory work outside of this RAP.

#### 11.8.8. Suppressive activity of regulatory cells

The list of analytes below will be listed only. PARAM/PARAMCD will be created from LBTEST/LBTESTCD and the Stimulus (Treg:Teff) an Stimulus concentrations (e.g. 0:1) which are stored in SUPPLB.

| Lab Test<br>(LBTEST) | Lab Test<br>Code<br>(LBTESTCD) | Units | Derived | Details |
|---|---|---|---|---|
| Count | COUNT | CPM | | |
| Percentage suppression | PCTSUPP | % | | |

The following stimulus will be used (stored in SUPPLB):

Treg:Teff

The following stimulus concentrations will be used (stored in SUPPLB):

- 0:1
- 1:1
- 1:2
- 1:4

### 11.8.9. Number of digits for display of biomarker data

To ensure that the outputs are readable, if the maximum value of the derived variable in the units given in this RAP is < 0.0001 both unit and values may be multiplied with  $10^3$ n (n being an integer) so that the maximum value is  $\ge 0.0001$ .

Otherwise, the following rules will apply:

- All individual continuous and count data will be displayed with three significant digits. Summary statistics will follow the normal IDSL rules, e.g. the mean will be presented with four significant digits.
- The display of percentages variable will depend on the median percentage across all treatments and time points, in the following manner:
  - The number of decimal points will be chosen so that the median as an individual value would be presented with three significant digits (e.g. if the median 20.5% all individual percentages should be displayed with one decimal place).
  - o Normal rules for derived summary statistics apply.
  - Any percentage larger than zero which would be displayed as zero according to the above rules will instead be displayed as "<X", where X is the smallest non-zero percentage that can be displayed.

# 11.9. Appendix 9: Abbreviations & Trademarks

# 11.9.1. Abbreviations

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CRS | Cytokine Release Syndrome |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| ECG | Electrocardiogram |
| EBV | Epstein-Barr virus |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| INS | Insulin |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMTT | Mixed Meal Tolerance Test |
| MMRM | Mixed Model Repeated Measures |
| PBMC | Peripheral Blood Mononuclear Cells |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| ULQ | Upper Limit of quantification |


OTX116505

| Abbreviation | Description |
|--------------|-----------------------|
| ULN | Upper Limit of Normal |

#### 11.9.2. Trademarks

| Trad | emarks of<br>Group | f the GI<br>of Com | thKline |
|------|--------------------|--------------------|---------|

| | lemarks not owned by the<br>nithKline Group of Companies |
|----------|----------------------------------------------------------|
| SAS | |
| SAS/STA | T |
| WinNonli | n |
| Spotfire | |

## 11.10. Appendix 10: List of Data Displays

## 11.10.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|--------------|
| Study Population | 1.01 to 1.XX | N/A |
| Safety | 2.01 to 2.XX | 2.01 to 2.XX |
| Efficacy | 3.01 to 3.XX | 3.01 to 3.XX |
| Pharmacodynamic | 4.01 to 4.XX | 4.01 to 4.XX |
| Biomarker | 5.01 to 5.XX | 5.01 to 5.XX |
| Pharmacokinetic | 6.01 to 6.XX | 6.01 to 6.XX |
| Section | List | ings |
| ICH Listings | 1 to XX | |
| Other Listings | XX+1 to ZZ | |

## 11.10.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 11: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-----------------|---------|---------|----------|
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Pharmacodynamic | PD_Fn | PD_Tn | PD_Ln |
| Biomarker | BIO_Fn | BIO_Tn | BIO_Ln |
| Listings | | | OTHER_Ln |

#### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

# 11.10.3. Deliverable [Priority]

The details provide abbreviations for the 'Delivery Priority' for the various reporting efforts for which displays will be generated.

| Abbreviation | Reporting Effort |
|--------------|----------------------------------------------|
| FA (SAC) | Final Analysis Statistical Analysis Complete |

# 11.10.4. Study Population Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Subject | Disposition | | | 1 | 1 |
| 1.01. | Enrolled | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | Programmer to update primary reason for withdrawal to be study specific. | FA (SAC) |
| 1.02. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | | FA (SAC) |
| 1.03. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | FA (SAC) |
| 1.04. | Enrolled | SP1 | Summary of Study Populations | | FA (SAC) |
| 1.05. | Safety | DV1 | Summary of Important Protocol Deviations | Generated, if data permits. As required, refer to PDMP. | FA (SAC) |
| 1.06. | Safety | SP3 | Summary of Exclusions from Per Protocol Population | | FA (SAC) |
| 1.07. | Safety | IE1 | Summary of Inclusion / Exclusion Criteria Deviations | | FA (SAC) |
| Demog | raphics | | * | 23 | 45 |
| 1.08. | Safety | DM1, DM5, DM<br>11 | Summary of Demographic Characteristics, Race and Racial Combinations and Age Ranges | Please combine shells in order DM1, DM5, DM 11. In addition those items please also add the categories for number of positive antibodies at screening (see Section 11.5.3) | FA (SAC) |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 1.09. | Safety | MH4 | Summary of Past and Current Medical Conditions | We only have current conditions, so need to display only those | FA (SAC) |
| Concor | mitant Medicati | ons | | | |
| 1.10. | Safety | CM7 | Summary of Concomitant Medications | Split as described in Section 11.3 | FA (SAC) |
| Exposi | ire | | | | |
| 1.11. | Safety | EX1 | Summary of Exposure to Study Drug | Also include daily infusion duration in hours for each dosing day | FA (SAC) |
## 11.10.5. Safety Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| AE | <del></del> | <del></del> | | * | A 40000 |
| 2.01. | Safety | AE13 | Adverse Event Overview | Split as described in Section 11.3 | FA (SAC) |
| 2.02. | Safety | AE15 | Summary of All Adverse Events by System Organ Class and Preferred Term | Split as described in Section 11.3 Add a "Any Event" category for each SOC even if not in shell | FA (SAC) |
| 2.03. | Safety | AE15 | Summary of Drug-Related Adverse Events | Split as described in Section 11.3 Add a "Any Event" category for each SOC even if not in shell | FA (SAC) |
| 2.04. | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term | Split as described in Section 11.3 | FA (SAC) |
| 2.05. | Safety | AE1 | Summary of AEs Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | Do not split this output by phase | FA (SAC) |
| 2.06. | Safety | AE5 | Summary of All Adverse Events by Maximum Grade by System<br>Organ Class and Preferred Term | Split as described in Section 11.3 | FA (SAC) |
| 2.07. | Safety | AE5 | Summary of Drug-Related Adverse Events by Maximum Grade by System Organ Class and Preferred Term | Split as described in Section 11.3 | FA (SAC) |

| 2.08. | Safety | AE15 | Summary of Adverse Events - Cytokine Release Syndrome Induced Symptoms | <ul> <li>Definition of Cytokine Release<br/>Syndrome in Section 11.5.3</li> <li>Overall only, not split by study<br/>phase.</li> </ul> | FA (SAC) |
|---|---|---|---|---|---|
| Epstein | -Barr Virus | | | , | |
| 2.09. | Safety | AE15 | Summary of Adverse Events Considered to be Potentially Associated with EBV Reactivation | Clinical Symptoms of Mononucleosis AE Terms to include are in Section 11.5.3 Overall only not split by study phase. | FA (SAC) |
| 2.10. | Safety | Non-Standard<br>SAFE_T3 | Summary of categorical values of Epstein-Barr Virus (Serology: IgG & IgM) | Categories (negative, positive) to be derived from absolute values according to a worst case approach as described in Section 11.5.3 | FA (SAC) |
| 2.11. | Safety | Non-Standard<br>SAFE_T2 | Summary of Epstein-Barr Viral Load (PCR) | Geometric Means | FA (SAC) |
| 2.12. | Safety | Non-Standard<br>SAFE_T4 | Categorical Summary of Epstein-Barr Viral Load (PCR) | | FA (SAC) |

| 2.13. | Safety | LB1 | Summary of Laboratory Values | <ul> <li>Order parameters<br/>alphabetically.</li> <li>BY Labtype (1. Chemistry, 2.<br/>Haematology)</li> </ul> | FA (SAC) |
|---|---|---|---|---|---|
| 2.14. | Safety | LB1 | Summary of Laboratory Changes from Baseline | <ul> <li>Order parameters<br/>alphabetically</li> <li>BY Labtype (1. Chemistry, 2.<br/>Haematology)</li> </ul> | FA (SAC) |
| 2.15. | Safety | LB15 | Summary of Worst Case Laboratory Results Relative to Normal Range Post-Baseline Relative to Baseline | <ul> <li>Order parameters<br/>alphabetically</li> <li>BY Labtype (1. Chemistry, 2.<br/>Haematology)</li> </ul> | FA (SAC) |
| Electro | cardiograms | | | | |
| 2.16. | Safety | EG1 | Summary of ECG Findings | | FA (SAC) |
| 2.17. | Safety | EG2 | Summary of Change from Baseline in ECG Values | | FA (SAC) |
| 2.18. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | | FA (SAC) |
| 2.19. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | | FA (SAC) |
| Vital Si | gns | | | | |
| 2.20. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | FA (SAC) |
| 2.21. | Safety | VS7 | Summary of Worst Case Vital Sign Results Relative to Potential Clinical Importance (PCI) Criteria Post-Baseline Relative to Baseline | | FA (SAC) |

| Immuno | Immunogenicity | | | | |
|---|---|---|---|---|---|
| 2.22. | Safety | Non-Standard<br>EFF_T4 | Summary of Immunogenicity | With positive instead of responder | FA (SAC) |

## 11.10.6. Safety Figures

| Safety | : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL No. /<br>E.G. Shell | Title | Programming Notes | Delivery<br>Priority |
| Labs | × = | )A | | | |
| 2.01 | Safety | SAF_F1 | Individual Subject Plot - Hematology & Clinical Chemistry<br>Selected Parameters | | FA (SAC) |
| Epstei | n-Barr Virus V | iral Load | | | |
| 2.02 | Safety | EFF_F2<br>(with<br>different<br>error bars,<br>see notes) | Geometric Mean (+/- CV%): Epstein-Barr Virus Viral Load | <ul> <li>X-axis: time</li> <li>Y-Axis: Geometric Mean Load (semi-log)</li> <li>Show error bars at (1+CV%) * GeoMean and GeoMean/(1+CV%)</li> <li>Line by group</li> </ul> | FA (SAC) |

## 11.10.7. Efficacy Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
|---|---|---|---|---|---|
| Mixed I | Meal Tolerance | Test : Weighted N | Mean AUC(0-120 mins) C-Peptide & Glucose | | |
| 3.01. | ITT<br>(Treated) | Non-Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline) : C-Peptide & Glucose Weighted Mean AUC(0-120 mins) from Mixed Meal Tolerance Test | | FA (SAC) |
| 3.02. | ITT<br>(Treated) | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline : C-Peptide & Glucose Weighted Mean AUC(0-120 mins) from Mixed Meal Tolerance Test | Include related estimated<br>LSMeans and treatment<br>differences. | FA (SAC) |
| 3.03. | Fully<br>Treated | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline : C-Peptide & Glucose Weighted Mean AUC(0-120 mins) from Mixed Meal Tolerance Test | Include related estimated LSMeans and treatment differences. | FA (SAC) |

| 2.04 | ITT | Non-Standard | Summary Statistics (Absolute and Change from Baseline): | | FA (SAC) |
|---|---|---|---|---|---|
| 3.04. | (Treated) | EFF_T1 | C-Peptide and Glucose Weighted Mean AUCs (60-140 mins) from Hyperglycemic Clamp Test | | |
| 3.05. | ITT<br>(Treated) | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline : C-Peptide and Glucose Weighted Mean AUCs (60-140 mins) from Hyperglycemic Clamp Test | Include related estimated LSMeans and treatment differences. | FA (SAC) |
| 3.06. | Fully<br>Treated | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline : C-Peptide and Glucose Weighted Mean AUCs (60-140 mins) from Hyperglycemic Clamp Test | Include related estimated LSMeans and treatment differences. | FA (SAC) |
| CLAMP | (Insulin Sensi | tivity Index) | | | |
| 3.07. | ITT<br>(Treated) | Non-Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline) : Insulin Sensitivity Index from Hyperglycemic Clamp Test | | FA (SAC) |
| 3.08. | ITT<br>(Treated) | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline : Insulin Sensitivity Index from Hyperglycemic Clamp Test | Include related estimated LSMeans and treatment differences. | FA (SAC) |
| Mean D | aily Insulin Us | 9 | | | |
| 3.09. | ITT<br>(Treated) | Non-Standard<br>EFF_T1 | Summary Statistics: (Absolute, Change from Baseline and Percentage Change from Baseline): Mean Daily Insulin Use | Please add percentage change<br>from baseline to the shell (as BY) | FA (SAC) |
| 3.10. | ITT<br>(Treated) | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline : Mean Daily Insulin Use | Include related estimated LSMeans and treatment differences. | FA (SAC) |
| %HbA1 | С | W. 2 | | * | |

| 3.11. | ITT<br>(Treated) | Non-Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline) : %HbA1c | | FA (SAC) |
|---|---|---|---|---|---|
| 3.12. | ITT<br>(Treated) | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline: %HbA1c | Include related estimated LSMeans and treatment differences. | FA (SAC) |
| Body V | Veight | | | | |
| 3.13. | ITT<br>(Treated) | Non-Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline) : Body Weight | | FA (SAC) |
| 3.14. | ITT<br>(Treated) | Non-Standard<br>EFF_T2 | Summary of Statistical Analysis (MMRM) Results of Change from Baseline: Body Weight | Include related estimated LSMeans and treatment differences. | FA (SAC) |
| Hypogl | ycemic & Hype | rglycemic Events | | | |
| 3.15. | ITT<br>(Treated) | Non-Standard<br>EFF_T3 | Summary of Hypoglycaemic & Hyperglycaemic Events by Intensity, SAE Status, Relationship to Investigational Product and Withdrawal Status | | FA (SAC) |
| Respon | nder Status | ng p | | | •<br>• |
| 3.16. | ITT<br>(Treated) | Non-Standard<br>EFF_T4 | Number and Percent of Subjects Meeting Definition of Glycemic Responder | Include Partial Remission Status and Hba1c responder status | FA (SAC) |
| 3.17. | ITT<br>(Treated) | Non-Standard<br>EFF_T4 | Number and Percent of Subjects Meeting Definition of C-Peptide Responder | | FA (SAC) |

## 11.10.8. Efficacy Figures

| Efficac | y Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL No. /<br>E.G. Shell | Title | Programming Notes | Deliverable<br>Priority |
| Mixed I | Meal Tolerance | Test : Weighted N | lean AUC(0-120 mins) C-Peptide & Glucose | | |
| 3.01 | ITT<br>(Treated) | Non- Standard<br>EFF_F1 | Model Adjusted Mean (+/- SE) Change from Baseline<br>Plot: C-Peptide & Glucose Weighted Mean AUC(0-<br>120 mins) from Mixed Meal Tolerance Test | By : Parameter X-Axis : Continuous scale for visit (months) Y-Axis : Mean (+/- SD) Chg from BL : Continuous scale for visit (moths) Legend : Treatment | FA (SAC) |
| Clamp | (Hyperglycaem | ic Phase) : Weigh | ted Mean AUCs (60-140 & 0-140 mins) C-Peptide & GI | ucose | 9 |
| 3.02 | ITT<br>(Treated) | Non- Standard<br>EFF_F1 | Model Adjusted Mean (+/- SE) Change from Baseline Plot: C-Peptide Weighted Mean AUCs (60-140 mins) from Hyperglycaemic Clamp Test | As Figure 3.01, adapted accordingly to the data | FA (SAC) |
| Mean D | aily Insulin Use | | | | |
| 3.03 | ITT<br>(Treated) | Non-Standard<br>EFF_F1 | Model Adjusted Mean (+/- SE) Change from Baseline Plot : Mean Daily Insulin Use | As Figure 3.01, adapted accordingly to the data | FA (SAC) |
| %HbA1 | С | | | | |
| 3.04 | ITT<br>(Treated) | Non- Standard<br>EFF_F1 | Model Adjusted Mean (+/- SE) Change from Baseline Plot : %HbA1c | As Figure 3.01, adapted accordingly to the data | FA (SAC) |
| Hyperg | lycemic and hy | poglycemic event | s by month | | |

| Efficac | Efficacy Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL No. /<br>E.G. Shell | Title | Programming Notes | Deliverable<br>Priority |
| 3.05 | ITT<br>(Treated) | EFF_F2 | Mean (+/- SE) Number of hyperglycemic and hypoglycemic events by month | | FA (SAC) |

## 11.10.9. Pharmacodynamic Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Pharma | acodynamic | | | · | |
| 4.01. | Safety | Non- Standard<br>PD_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Target Engagement | For parameters with imputation please also include no. of subjects with LLQs & ULQ. Include the parameters to be summarized from 11.5.5 and also show the two derived % Target Engagement variables | FA (SAC) |

# 11.10.10. Pharmacodynamic Figures

| Pharma | Pharmacodynamic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | codynamic | | 5)<br> | | |
| 4.01. | Fully<br>Treated | Non- Standard<br>EFF_F1 | Mean (+/- SE) Change from Baseline in Target Engagement | Pages BY parameters, same as table. Lines by group. Please show same parameters as in Table 4.01. | FA (SAC) |

## 11.10.11. Biomarker Tables

| Biomar | Biomarker : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Biomar | ker | | | | |
| 5.01. | Fully<br>Treated | Non- Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Frequency and phenotype of lymphocyte subsets by flow<br>cytometry | | FA (SAC) |
| 5.02. | Fully<br>Treated | EFF_T5 | Summary Statistics (Absolute and Change from Baseline):<br>Frequency and phenotype of lymphocyte subsets by flow<br>cytometry by C-Peptide Response | | FA (SAC) |
| 5.03. | Multimer<br>Analyses | Non- Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Frequency and phenotype of HLA-A2-resticted EBV-specific<br>CD8+ T cells by multimer analysis | | FA (SAC) |
| 5.04. | Fully<br>Treated | Non- Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline):<br>Quantification of serum cytokines and soluble cytokine receptors | | FA (SAC) |
| 5.05. | Fully<br>Treated | Non- Standard<br>EFF_T1 | Summary Statistics (Absolute and Change from Baseline): TCR deep sequencing | | FA (SAC) |

# 11.10.12. Biomarker Figures

| Biomarl | ker : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Biomarl | ker | | | | · |
| 5.01. | Fully Treated | EFF_F3 | Mean (+/- SE) Change from Baseline in Frequency and phenotype of lymphocyte subsets by flow cytometry by C-Peptide Response | | FA (SAC) |

## 11.10.13. Pharmacokinetic Tables

| Pharma | cokinetic : Tab | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 6.01 | Fully<br>Treated | PK01 | Summary of Free Serum Otelixizumab Concentration-Time Data by Treatment | | FA (SAC) |

## 11.10.14. Pharmacokinetic Figures

| Pharma | acokinetic : Fig | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Cor | centration | A | | | |
| 6.01 | Fully<br>Treated | PK16a | Individual Free Serum Otelixizumab Concentration-Time Plots (Linear and Semi-Log) by Subject | | FA (SAC) |
| 6.02 | Fully<br>Treated | PK17 | Mean Free Serum Otelixizumab Concentration-Time Plots by<br>Treatment (Linear and Semi-Log) | Use geometric mean for semi-log scale | FA (SAC) |
| 6.03 | Fully<br>Treated | PK18 | Median Free Serum Otelixizumab Concentration-Time Plots by Treatment (Linear and Semi-Log) | | FA (SAC) |

## 11.10.15. ICH Listings

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | misation | | | | |
| 01. | Randomised | TA1 | Listing of Randomised and Actual Treatments | | FA (SAC) |
| Subjec | t Disposition | | | | |
| 02. | Enrolled | ES2 | Listing of Reasons for Study Withdrawal | | FA (SAC) |
| 03. | Safety | SD2 | Listing of Reasons for Study Treatment Discontinuation | | FA (SAC) |
| 04. | Enrolled | DV2 | Listing of Important Protocol Deviations | | FA (SAC) |
| 05. | Enrolled | SP3 | Listing of Exclusions from Any Population | | FA (SAC) |
| 06. | Screened | ES7 | Listing of Reason for Screen Failure | | FA (SAC) |
| 07. | Enrolled | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | FA (SAC) |
| Exposi | ure | at. | | | |
| 08. | Safety | EX3 | Listing of Exposure Data | <ul> <li>List each infusion, we will give duration in minutes (end of infusion – start of infusion).</li> <li>We can omit Dosing</li> </ul> | FA (SAC) |
| Domos | ranhias | м. | | Frequency. | - |
| | raphics | D. C. | | Ī | E1 /515 |
| 09. | Safety | DM2 | Listing of Demographic Characteristics | | FA (SAC) |
| 10. | Safety | DM9 | Listing of Race | | FA (SAC) |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 11. | Safety | Non-Standard<br>OTHER_L10 | Listing of Family History of Cardiovascular Risk | | FA (SAC) |
| 12. | Safety | Non-Standard<br>OTHER_L11 | Listing of Substance Use | | FA (SAC) |
| Conme | ds | | | | |
| 13. | Safety | CM3 | Listing of Concomitant Medications | Include ATC/Ingredient | FA (SAC) |
| 14. | Safety | Non-Standard<br>OTHER_L6 | Listing of Insulin Use | CMCAT = DAILY INSULIN USE | FA (SAC) |
| AE | J. | | | | |
| 15. | Safety | AE8 | Listing of All Adverse Events | | FA (SAC) |
| 16. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | FA (SAC) |
| 17. | Safety | AE8CPA | Listing of Serious Adverse Events | | FA (SAC) |
| 18. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | FA (SAC) |
| 19. | Safety | AE8 | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | FA (SAC) |
| 20. | Safety | AE2 | Relationship of Adverse Event SOCs, PTs, and Verbatim Text | | FA (SAC) |
| 21. | Safety | AE8 | Listing of All Adverse Events - Cytokine Release Syndrome Induced Symptoms | See Section 11.5.3 for definition | FA (SAC) |

| ICH : L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 22. | Safety | AE8 | Listing of All Adverse Events – Considered Potentially Associated with EBV Reactivation | See Section 11.5.3 for definition | FA (SAC) |
| 23. | Safety | OTHER_L12 | Listing of Epstein-Barr Virus Serology: IgG & IgM and Viral Load: PCR | Please include the following:<br>EBCIGGAS, EBVMSOS, EBCIGGAB,<br>EBVMABZ, EBCIGMAB, EBVDNA | FA (SAC) |
| LABS | | 7.<br>C | | | · · |
| 24. | Safety | LB5 | Listing of All Haematology Laboratory Data for Subjects with Abnormalities of Potential Clinical Importance | | FA (SAC) |
| 25. | Safety | LB14 | Listing of Haematology Laboratory Data with Character Results | | FA (SAC) |
| 26. | Safety | LB5 | Listing of All Clinical Chemistry Laboratory Data for Subjects with Abnormalities of Potential Clinical Importance | | FA (SAC) |
| 27. | Safety | LB14 | Listing of Clinical Chemistry Laboratory Data with Character Results | | FA (SAC) |
| 28. | Safety | LB5 | Listing of All Serology Data | | FA (SAC) |
| 29. | Safety | LB14 | Listing of Serology Data with Character Results | | FA (SAC) |
| ECG's | | l. | | | |
| 30. | Safety | EG3 | Listing of ECG Values of Potential Clinical Importance | | FA (SAC) |
| 31. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | Including change from Baseline | FA (SAC) |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 32. | Safety | EG5 | Listing of Abnormal ECG Findings | | FA (SAC) |
| Vital Si | gns | Į. | | <del>.</del> | |
| 33. | Safety | VS4 | Listing of Vital Signs of Potential Clinical Importance | | FA (SAC) |
| 34. | Safety | VS4 | Listing of All Vital Signs for Subjects with Values of Potential Clinical Importance | | FA (SAC) |
| Pharma | acokinetics | 37 A | | * | * |
| 35. | Safety | PK07 | Listing of free serum concentration-Time Data | | FA (SAC) |

OTX116505

## 11.10.16. Non-ICH Listings

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study F | opulation, Saf | ety and Efficacy | | | |
| 36. | Safety | CP_ML1 p | Listing of Dosing Times, Meal Start and End Times on Fed Treatment Days | Classify as Safety for HARP/SAFIRE | FA (SAC) |
| 37. | Safety | Non-Standard<br>Other_L4 | Listing of Auto-Antibody Results | Classify as Study Population for HARP/SAFIRE | FA (SAC) |
| 38. | Safety | Non-Standard<br>Other_L3 | Listing of Immunogenicity Results | Classify as Safety for HARP/SAFIRE | FA (SAC) |
| 39. | Safety | Non-Standard<br>Other_L1 | Listing of C-Peptide & Glucose from Mixed Meal Test | <ul> <li>List by Parameter</li> <li>Absolute and change from baseline result to be presented.</li> </ul> | FA (SAC) |
| 40. | Safety | Non-Standard<br>Other_L2 | Listing of C-Peptide & Glucose from Mixed Meal Test: Derived Parameters | <ul> <li>List by Parameter</li> <li>Absolute and change from baseline result to be presented.</li> <li>Also include C-peptide response</li> </ul> | FA (SAC) |
| 41. | Safety | Non-Standard<br>Other_L8 | Listing of C-Peptide & Glucose from Clamp | List by Parameter Absolute and change from baseline result to be presented. | FA (SAC) |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 42. | Safety | Non-Standard<br>Other_L9 | Listing of C-Peptide & Glucose from Clamp : Derived Parameters | <ul> <li>List by Parameter</li> <li>Absolute and change from baseline result to be presented.</li> </ul> | FA (SAC) |
| 43. | Safety | Non-Standard<br>Other_L1 | Listing of Insulin Sensitivity Index (Hyperglycemic Clamp), Mean Daily Insulin Usage and %HbA1c | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. Include glycemic response variables | FA (SAC) |
| 44. | Safety | Non-Standard<br>Other_L5 | Listing of Hypoglycemic & Hyperglycemic Event Rates | | FA (SAC) |
| 45. | Safety | Non-Standard<br>Other_L7 | Cardiovascular Events | Classify as Safety for HARP/SAFIRE | FA (SAC) |
| Pharma | codynamics | · | | | |
| 46. | Safety | Non-Standard<br>Other_L1 | Listing of Pharmacodynamics including Target Engagement | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. | FA (SAC) |
| Biomar | kers | | | от опаропи. | |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 47. | ITT<br>(Treated) | Non-Standard<br>Other_L1 | Listing of frequency and phenotype of lymphocyte subsets by flow cytometry | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. | FA (SAC) |
| 48. | ITT<br>(Treated) | Non-Standard<br>Other_L1 | Listing of frequency of FoxP3 regulatory cells and TH17 cells by epigenetic quantification | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. | FA (SAC) |
| 49. | Multimer<br>Analyses | Non-Standard<br>Other_L1 | Listing of frequency and phenotype of HLA-A2-resticted antigen-<br>specific CD8+ T cells by multimer analysis | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. | FA (SAC) |
| 50. | ITT<br>(Treated) | Non-Standard<br>Other_L1 | Listing of frequency of interferon-gamma-secreting antigen-<br>reactive cells by ELISPOT | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. | FA (SAC) |
| 51. | ITT<br>(Treated) | Non-Standard<br>Other_L1 | Listing of quantification of serum cytokines and soluble cytokine receptors | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. | FA (SAC) |
| 52. | ITT<br>(Treated) | Non-Standard<br>Other_L1 | Listing of TCR deep sequencing results | Absolute and change from baseline result to be presented. Example Other_L1 modified based on endpoint. | FA (SAC) |

| Non-IC | H : Listings | | | | |
|---|---|---|---|---|---|
| No. Population | | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority]<br>FA (SAC) |
| 53. | ITT<br>(Treated) | Listing of suppressive activity of regulatory cells | | <ul> <li>Absolute and change from<br/>baseline result to be presented.</li> <li>Example Other_L1 modified based<br/>on endpoint.</li> </ul> | |
| Statisti | cal Listings | | | | |
| 54. | ITT<br>(Treated) | SAS Output | Statistical Output for Statistical Analysis (MMRM) Results of Change from Baseline : C-Peptide & Glucose Weighted Mean AUC(0-120 mins) from Mixed Meal Tolerance Test | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots Also include a listing showing the p-values for the model selection approach described in Section 9.1.5.1 in the following format: Covariate Type III P-value BMI 0.XXXXX (from 1) BMI*trt 0.XXXXX (from 2) Show this for each covariate, but do not include tests for the other variables in the model | FA (SAC) |
| 55. | ITT<br>(Treated) | SAS Output | Statistical Output for Statistical Analysis (MMRM) Results of<br>Change from Baseline : C-Peptide Weighted Mean AUCs (60-<br>140 mins) from Hyperglycemic Clamp Test | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots | FA (SAC) |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 56. | Fully<br>Treated | SAS Output | Statistical Output for Statistical Analysis (MMRM) Results of Change from Baseline : C-Peptide & Glucose Weighted Mean AUC(0-120 mins) from Mixed Meal Tolerance Test | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots | FA (SAC) |
| 57. | Fully<br>Treated | SAS Output | Statistical Output for Statistical Analysis (MMRM) Results of Change from Baseline : C-Peptide Weighted Mean AUCs (60-140 mins) from Hyperglycemic Clamp Test | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots | FA (SAC) |
| 58. | ITT<br>(Treated) | SAS Output | Statistical Output for Statistical Analysis (MMRM) Results of Change from Baseline : Insulin Sensitivity Index from Hyperglycemic Clamp Test | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots | FA (SAC) |
| 59. | ITT<br>(Treated) | SAS Output | Statistical Output for Statistical Analysis (MMRM) Results of Change from Baseline : Mean Daily Insulin Use | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots | FA (SAC) |
| 60. | ITT<br>(Treated) | SAS Output | Statistical Output for Statistical Analysis (MMRM) Results of Change from Baseline: %HbA1c | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots | |
| 61. | ITT<br>(Treated) | SAS Output | Summary of Statistical Analysis (MMRM) Results of Change from Baseline: Body Weight | Please include standard SAS output, including estimation of variance components, model diagnostics and residual plots | |

# 11.11. Appendix 11: Example Mock Shells for Data Displays


Protocol : OTX116505 Population : Safety

Figure X.XX

Model Adjusted Mean (95% CI) Change from Baseline Plot: C-Peptide & Glucose Weighted Mean AUC(0-120 mins) from Mixed Meal Tolerance Test



Programming Notes: [1] Include C-Pe

[1] Include C-Peptide and Glucose.

[2] Use OTX instead of OTE for treatment labels.

OTX116505

[3] An OTX 36 mg will not be included in the data (not dosed)


Protocol: OTX116505 Population: Safety

Figure X.XX

Mean (+/- SE) Number of hyperglycemic and hypoglycemic events by month



Programming Notes: [1] Example only; actual event rates are not assumed to stay constant over month.

OTX116505


Protocol: OTX116505 Population : Safety

Figure X.XX

Mean (+/- SE) Change from Baseline in Frequency and phenotype of lymphocyte subsets by flow cytometry by C-Peptide Response

| Programming Notes : | Similar to EFF_F1, but with: |
|---|---|
| | [1] Line by C-Peptide Responder Status [2] Panel by treatment |

Page 1 of X Example : SAF\_F1

Protocol: OTX116505 Population : Safety

Figure X.XX Individual Subject Plot - Hematology & Clinical Chemistry Selected Parameters

Category: Hematology; Parameter: Leukocytes (GI/L) Treatment: Placebo; Time Span: All data



Programming Notes: Similar to EFF\_F1, but with:

OTX116505

- [1] Line by C-Peptide Responder Status [2] Panel by treatment

OTX116505


**Example : SAFE\_T1**Table SAFE\_T1 has been deprecated and will not be used.

OTX116505

Example : SAFE\_T2 Protocol: OTX116505


Population : Safety

#### Table X.XX

Summary (Absolute and Change from Baseline) of Epstein-Barr Virus (Viral Load: PCR)

Summary: Absolute

| Treatment | Time | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | 95% Confidence Interval for | | | | | | | |
| | | N | n | Mean/Geo. Mean | Geometric Mean | CVb% | Min | Median | Max |
| Placebo | X | х | x | xxx.x/xxx.x | xxx.x; xxx.x | XX% | XXX | xxx | Xxx |
| | X | х | x | xxx.x/xxx.x | xxx.x; xxx.x | XX% | xxx | xxx | Xxx |
| | X | X | X | xxx.x/xxx.x | XXX.X; XXX.X | XX% | XXX | XXX | Xxx |
| | | 0.00 | | | * (*) | | * | >• | (*) |
| OTX 9 mg | Χ | х | х | xxx.x/xxx.x | xxx.x; xxx.x | XX% | XXX | XXX | Xxx |
| • | X | x | x | xxx.x/xxx.x | xxx.x; xxx.x | XX% | xxx | xxx | Xxx |
| | X | x | x | xxx.x/xxx.x | xxx.x; xxx.x | XX% | xxx | xxx | Xxx |
| | * | | | ¥ | ¥ (¥) | | ¥ | 2 | |
| | * | | | \$ <b>.0</b> \$ | | 236 | * | • | |

Continue for other doses

[1] For applicable endpoints, include parameter as either a BY parameter or as first column in the table [2] CVb%: calculate SD on log scale and then CVb% = 100\*sqrt(exp(SD^2)-1)) with SD being the SD on log scale. Programming Notes:

OTX116505


Example : SAFE\_T2 (Continued)

Protocol : OTX116505 Population : Safety

Table X.XX

Summary (Absolute and Change from Baseline) of Epstein-Barr Virus (Viral Load: PCR)

Summary: Change from Baseline

ETC

Programming Notes: [1] For applicable endpoints, include parameter as either a BY parameter or as first column in the table
**Example : SAFE\_T3**Protocol : OTX116505
Population : Safety


 Table X.XX

 Summary of Categorical values of Epstein-Barr Virus (Serology:lgG & lgM)

| | | | | | | | Number of | of Subjects (%) | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Absolut | e Values | Change from Baseline | | | |
| Parameter | Visit | Treatment | N | n | Positive | Negative | Positive-<br>Positive | Positive-<br>Negative | Negative-<br>Positive | Negative-<br>Negative |
| Epstein-<br>Barr IgG<br>Antibody | Screening | Placebo | XX | XX | XX (%) | XX (%) | | | | |
| | | OTX 9 mg | XX | XX | XX (%) | XX (%) | | | | |
| | | OTX 18 mg | XX | XX | XX (%) | XX (%) | | | | |
| | | OTX 27 mg | XX | XX | XX (%) | XX (%) | | | | |
| | Day -1 | Placebo | XX | XX | XX (%) | XX (%) | | | | |
| | | OTX 9 mg | XX | XX | XX (%) | XX (%) | | | | |
| | | OTX 18 mg | XX | XX | XX (%) | XX (%) | | | | |
| | | OTX 27 mg | XX | XX | XX (%) | XX (%) | | | | |
| | Day 6 | Placebo | XX | XX | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | OTX 9 mg | XX | XX | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | OTX 18 mg | XX | XX | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |
| | | OTX 27 mg | XX | XX | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) | XX (%) |

OTX116505

Example : SAFE\_T4

Protocol : OTX116505 Population : Safety Page 1 of X

Table X.XX

Categorical Summary of Epstein-Barr Virus (Viral Load: PCR)

Unit: copies/10^6PBM cells

| Treatment | Visit | | | | Number of | Subjects (%) | |
|---|---|---|---|---|---|---|---|
| | | N | n | 0-1000 | >1000-10000 | >10000-100000 | >100000 |
| Placebo | Х | x | | XX (%) | XX (%) | XX (%) | XX (%) |
| | X | x | | XX (%) | XX (%) | XX (%) | XX (%) |
| | X | x | | XX (%) | XX (%) | XX (%) | XX (%) |
| | ¥ | 130 | | | | | |
| OTX 9 mg | X | x | | XX (%) | XX (%) | XX (%) | XX (%) |
| | X | X | | XX (%) | XX (%) | XX (%) | XX (%) |
| | Χ | X | | XX (%) | XX (%) | XX (%) | XX (%) |
| | | • | | | i i | ************************************** | 8 |
| | * | ne | | 36 36 | 3*2 64 | | |

ETC

Programming Notes: [1] For applicable endpoints, include parameter as either a BY parameter or as first column in the table

OTX116505

Example : **EFF\_T1**Protocol : OTX116505

Population : Safety


#### Table X.XX

Summary Statistics (Absolute and Change from Baseline): C-Peptide & Glucose from Mixed Meal Tolerance Test

Parameter: C-peptide Weighted Mean AUC 0-120 mins (nmol/L)

| Treatment | N | Visit | Variable | n | Mean | 95% Confidence Interval | SD | Min | Median | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | Х | Screening | Abs. | Х | xxx.x | xxx.x, xxx.x | xx.xx | xxx | xxx | Xxx |
| | | Month 3 | Abs. | X | XXX.X | xxx.x, xxx.x xxx xxx xxx | Xxx | | | |
| | | XXXX | Chg. | X | XXX.X | xxx.x, xxx.x | xx.xx xxx xxx | Xxx | | |
| | | Month 6 | Abs. | X | XXX.X | XXX.X, XXX.X | xx.xx | XXX | XXX | Xxx |
| | | XXXX | Chg. | X | XXX.X | xxx.x, xxx.x | xx.xx | xxx | xxx | Xxx |
| | | XXXX | | X | XXX.X | XXX.X, XXX.X | xx.xx | XXX | xxx<br>xxx<br>xxx<br>xxx | Xxx |
| OTX 9 mg | | XXXX | | Х | XXX.X | xxx.x, xxx.x | xx.xx | XXX | XXX | Xxx |
| | | XXXX | | X | xxx.x | xxx.x, xxx.x | XX.XX | XXX | XXX | Xxx |
| | | XXXX | | X | XXX.X | XXX.X, XXX.X | XX.XX | XXX | XXX | Xxx |
| * | | | | | *: | | | (6) | | |

Programming Notes: [1] For applicable endpoints, include parameter as either a BY parameter or as first column in the table

OTX116505

Example : EFF\_T1 (Continued) Page 1 of X

Protocol : OTX116505 Population : Safety

#### Table X.XX

Summary Statistics (Absolute and Change from Baseline): C-Peptide & Glucose from Mixed Meal Tolerance Test

Summary: Change from Baseline

Please use same shell as for absolute values

| Programming Notes : | [1] For applicable endpoints, include parameter as either a BY parameter or as first column in the table |
|---|---|
| | [2] If later it is decided to use log-transformation instead, then please use SAFE T-2 as template for them. |
| | [3]: If not all columns fit on one page, please switch to PD_T1 instead. |

Example : EFF\_T2 Page 1 of X

Protocol : OTX116505 Population : Safety

#### Table X.XX

Summary of Statistical Analysis (MMRM) Results of Change from Baseline: C-Peptide & Glucose Weighted Mean AUC(0-120 mins) from Mixed Meal Tolerance Test

#### Parameter:

| Visit | Statistic | Placebo<br>N=xx | OTX 9 mg<br>N=xx | OTX 18 mg<br>N=xx | OTX 27 mg<br>N=xx |
|---|---|---|---|---|---|
| Month 3 | n(1) | xx | xx | xx | xx |
| | n(2) | xx | xx | xx | xx |
| | LS Mean | x.xx | x.xx | x.xx | x.xx |
| | LS Mean Change | x.xx | x.xx | x.xx | x.xx |
| | Standard Error | x.xxx | x.xxx | x.xxx | x.xxx |
| | Difference from Placebo | | x.xx | x.xx | x.xx |
| | 95% Confidence Interval | | x.xx - x.xx | x.xx - x.xx | x.xx - x.xx |
| | P-value | | 0.xxx | 0.xxx | 0.xxx |

| Footnotes : | n(1) = Number of subjects in analysis; n(2) = Number of subjects with data at that visit |
|---|---|
| | P-value tests the null hypothesis of no difference from placebo. |
| Programming Notes | Use three decimal places for p-values. Always use ceiling instead of rounding (i.e. show 0.0501 as 0.051 and not 0.050. If the p-value is smaller than 0.001 display as "< 0.001". |

Example : EFF\_T3 

Protocol: OTX116505 Population: Safety

### **Table X.XX**Summary of Hypoglycaemic & Hyperglycaemic Events and Event Rates

#### Hypoglycaemic Events

| | | Placebo<br>(N=xxx) | 8 | 16. | 9mg<br>(N=xxx) | |
|---|---|---|---|---|---|---|
| Time Period<br>Category | n (%) | Number of<br>Events /<br>Mean [1] | Time<br>Normalized<br>Number of<br>Events /<br>Mean [2] | n/N (%) | Number of<br>Events / Mean<br>[1] | Time Normalized<br>Number of<br>Events / Mean<br>[2] |
| Any Time Post-dose | | | | | | |
| Number of Subjects | X | | | X | | |
| Any Hypoglycemia | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx/xxx (xx%) | xxx / xx.x | xxx / xx.x |
| Hypoglycemia Grade 1 | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx/xxx (xx%) | xxx / xx.x | xxx / xx.x |
| Hypoglycemia Grade 2 | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx/xxx (xx%) | xxx / xx.x | xxx / xx.x |
| Hypoglycemia Grade 3 | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx/xxx (xx%) | xxx / xx.x | xxx / xx.x |
| <b>*</b> | | | | | | |
| Dosing Period | | | | | | |
| Number of Subjects | X | | | X | | |
| Any Hypoglycemia | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx (xx%) | xxx / xx.x | xxx / xx.x |
| Hypoglycemia Grade 1 | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx (xx%) | xxx / xx.x | xxx / xx.x |
| Hypoglycemia Grade 2 | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx (xx%) | xxx / xx.x | xxx / xx.x |
| Hypoglycemia Grade 3 | xxx (xx%) | xxx / xx.x | xxx / xx.x | xxx (xx%) | xxx / xx.x | xxx / xx.x |
| 90-35 500 F2<br>4-00- | | | | | | |

<sup>[1]</sup> Number of Events = the total number of events at each level of summarization. Mean = the average

OTX116505

number of events reported per subject.

[2] Normalized by dividing Number of Events by length of reporting period in month (1 month = 30 days). Mean = the average event rate reported by subject. Subjects are only included if they had both visits delimiting the reporting period.

| Programming Notes : | [1] Please show same categories as AE tables by grade: grades 1,2,3,4,5 as well as grade 3+4+5 and unknown (if any). |
|---|---|
| | [2] Continue with Post-dose up to Week 6 Visit, Post Week 6 Visit to Month 3 Visit, Post Month 3 Visit to Month 6 visit then similarly, 6-9, 9-12, 12-18, |
| | 18-24. Please continue with Hyperglycaemic events and update the footnote accordingly. Please use the Number of Subjects row in each column as |
| | the denominator for the percentages, not the overall N. |

Example : EFF\_T4 

Protocol : OTX116505 Population : Safety

 Table X.XX

 Number and Percent of Subjects Meeting Definition of Glycemic Responder

| | | | Pl | acebo | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Visit | Responder Status | N | XX= | OTX | 9 mg | OTX | 18 mg | OTX | 27 mg |
| Glycemic Response | Week 4 | Responders | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) |
| 9E3 | | Non-responders | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) |
| | | New responders | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) |
| | | Non-responders who were responders at previous visit | XX | (XX%) | XX | (XX%) | XX | (XX%) | XX | (XX%) |
| | Week X | *** | | | | | | | | |

Note: a subject is a glycemic responder, if he fulfils the following criteria:

<sup>1.</sup> HbA1c <= 7%

<sup>2.</sup> Mean daily insulin use < 0.5 units/kg/day.

OTX116505

Example : EFF\_T5

Protocol : OTX116505 Population : Safety Page 1 of X

#### Table X.XX

Summary Statistics (Absolute and Change from Baseline): Frequency and phenotype of lymphocyte subsets by flow cytometry by C-Peptide Response

Parameter: XXXXX (UNIT)

Summary: Absolute

| | | | cebo<br>=XX | | 9 mg<br>=XX | | 18 mg<br>≡XX | | 27 mg<br>=XX |
|---|---|---|---|---|---|---|---|---|---|
| | | Non- | | Non- | | Non- | | 74 4 10 0 T 17 T 17 T 17 T 17 T 17 T 17 T 17 | <b>-</b> 960-1500000- <b>3</b> 66700-2 |
| Visit | Statistic | responders | Responders | responders | Responders | responders | Responders | Non-responders | Responders |
| Screening | n | xx | xx | XX | XX | xx | XX | xx | xx |
| | Mean | XXX.X | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x | xxx.x |
| | 95%<br>Confidence<br>Interval | XXX.X; XXX.X | XXX.X; XXX.X | xxx.x;<br>xxx.x | xxx.x; xxx.x | xxx.x; xxx.x | XXX.X; XXX.X | xxx.x; xxx.x | XXX.X; XXX.X |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | xx.xx | XX.XX | XX.XX |
| | Min | XXX | XXX | XXX | XXX | XXX | XXX | xxx | xxx |
| | Median | XXX | XXX | XXX | XXX | XXX | xxx | xxx | xxx |
| | Max | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| ••• | (8.8.5) | | | | | | | | |
| | | 12 | | | | | | | |

ETC

| Programming Notes : | Footnotes: |
|---|---|
| | [1] A participant is considered a C-peptide responder if there is >-40% change from baseline in C-peptide MMTT Weighted Mean AUC (0-120) after 24 |
| 14 | months. |

OTX116505

[2] Subjects with missing responder status due to missing C-peptide at 24 months are not included in the table.

OTX116505

Example: PD\_T1
Protocol: OTX116505

Population : Safety


#### Table X.XX

Summary Statistics (Absolute and Change from Baseline): Target Engagement

Parameter: XXXXX

| Treatment | N | Visit, Time | Variable | n | Mean | 95% Confidence Interval | SD | Min | Median | Max |
|---|---|---|---|---|---|---|---|---|---|---|
| Placebo | Х | Day 1, 00:00 | Abs. | Х | XXX.X | xxx.x, xxx.x | xx.xx | XXX | xxx | Xxx |
| | | | Chg. | X | XXX.X | xxx.x, xxx.x | XX.XX | xxx | xxx | Xxx |

...

OTX 9 mg

x x x x x x

ETC

OTX116505

Example : OTHER\_L1

Protocol: OTX116505 Population : Safety


Listing XX
Listing of C-Peptide & Glucose from Mixed Meal Tolerance Test

Treatment:Placebo

| Inv./<br>Subj. | Age(yrs)/<br>Sex/<br>Race | Visit | Date/<br>Study Day | Planned/Actual<br>Relative<br>Time<br>(Mins) | Time<br>Sample<br>Taken | C-Peptide<br>(Units) | Glucose<br>(Units) |
|---|---|---|---|---|---|---|---|
| XXXXX/<br>XXX | XX/<br>Male/<br>White | XXXX | DDMMMYYYY / XX | X/X | HH:MM | XXX.XX | XXX.XX |
| | | | | X | HH:MM | XXX.XX | XXX.XX |
| | | | | X | HH:MM | XXX.XX | XXX.XX |
| | | | | X | HH:MM | XXX.XX | XXX.XX |
| | | | | X | HH:MM | XXX.XX | XXX.XX |
| | | XXXX | DDMMMYYYY | Х | HH:MM | XXX.XX | XXX.XX |
| | | | | X | HH:MM | XXX.XX | XXX.XX |
| | | | | X | HH:MM | XXX.XX | XXX.XX |

[1] As required to be modified based on data and any applicable IDSL standard principles for listings Programming Notes :

OTX116505

Example : OTHER\_L2

Protocol : OTX116505 Population : Safety Page 1 of X

#### Listing XX

Listing of C-Peptide & Glucose from Mixed Meal Test: Derived Parameters

Treatment: Placebo

| Inv./Subj. | Age(yrs)/<br>Sex/<br>Race | Analyte | Visit | Date/Study Day | Time Int. For<br>Derivation<br>(Mins) | Weighted<br>Mean<br>AUC(0-120M)<br>Results | Change<br>from Baseline<br>Weighted Mean<br>AUC(0-120M) |
|---|---|---|---|---|---|---|---|
| XXXXX/ XXX | XX/<br>Male/ | XXXXX | XXXX | DDMMMYYYY / XX | XXX | X.XXX | X.XXX |
| | White | | | | | | |
| | | | XXXX | | XXX | X.XXX | X.XXX |
| | | | XXXX | | XXX | X.XXX | X.XXX |
| | | | XXXX | | XXX | X.XXX | X.XXX |
| | | xxxxx | XXXX | | | X.XXX | X.XXX |
| | | | XXXX | | | X.XXX | X.XXX |
| | | | XXXX | | | X.XXX | X.XXX |
| | | | XXXX | | | X.XXX | X.XXX |

Programming Notes: [1] As required to be modified based on data and any applicable IDSL standard principles for listings

OTX116505


Protocol : OTX116505 Population : Safety

# Listing XX Listing of Immunogenicity Results

#### Treatment: Placebo

| Inv./<br>Subj. | Age(yrs)/<br>Sex/<br>Race | Visit | Date/Time sample<br>Taken | Screening<br>Result | Confirmation<br>Result | Titer |
|---|---|---|---|---|---|---|
| Xxxx/<br>xxx | XX/<br>Male/<br>White | Day -1 | DDMMMYYYY/Hh:mm | Positive | Positive | Х |

| 2 | |
|---|---|
| Programming Notes : | [1] As required to be modified based on data and any applicable IDSL standard principles for listings |

OTX116505

Example : OTHER\_L4

<u>\_</u>\_\_\_\_4


Protocol : OTX116505 Population : Safety

# **Listing XX**Listing of Auto-Antibody Results

#### Treatment:Placebo

| Inv./<br>Subj. | Age(yrs)/<br>Sex/<br>Race | Visit | Date | Study<br>Day | Time | Result | Unified<br>Classifica<br>tion |
|---|---|---|---|---|---|---|---|
| Xxxx/<br>xxx | 27/<br>Male/<br>White | Screening | DDMMMYYYY | XX | XX:XX | xxxx | XXXX |

| <u> </u> | |
|---|---|
| Programming Notes : | [1] As required to be modified based on data and any applicable IDSL standard principles for listings |

OTX116505


Protocol : OTX116505 Population : Safety

# Listing XX Listing of Hypoglycemic & Hyperglycemic Event Rates

Treatment: Placebo

| Inv./<br>Subj. | Age(yrs)/<br>Sex/<br>Race | Event Type | Reporting<br>Period | Number<br>of<br>Events | Start/End Date<br>of Reporting<br>Period | Duration of reporting period (months) | Event Rate (1/month) |
|---|---|---|---|---|---|---|---|
| Xxxx/<br>xxx | 27/<br>Male/<br>White | Hypoglycemic | Overall (up to 24 months visit) | XXXX | DDMMMYYYY/<br>DDMMMYYYY | XXX | XXXX |
| | | | Dosing<br>Period | XXXX | DDMMMYYYY/<br>DDMMMYYYY | XXXX | XXXX |
| | | | Post Dosing<br>Period up<br>to 6 weeks | XXXX | DDMMMYYYY/<br>DDMMMYYYY | XXXX | XXXX |
| | | | 6 weeks to<br>3 months | XXXX | DDMMMYYYY/ | | |

| Footnotes: | For the purpose of this listing one month is assumed to have 30 days. Duration of period and event rate will only be calculated if the visit at the end of the reporting period took place. |
|---|---|
| Programming Notes : | [1] As required to be modified based on data and any applicable IDSL standard principles for listings |

OTX116505

Example : OTHER\_L6

Protocol : OTX116505 Population : Safety Page 1 of X

Listing XX
Listing of Insulin Use

Treatment: Placebo

| Inv./<br>Subj. | Age(yrs)/<br>Sex/<br>Race | Study Day | Date/Time | Reported<br>Name/<br>Standardized<br>Name | Dose | Unit | Last<br>Recorded<br>Weight Prior<br>to Intake<br>(kg) | Standardized<br>Dose<br>(IU/kg) |
|---|---|---|---|---|---|---|---|---|
| Xxxx/<br>xxx | 27/<br>Male/<br>White | xxxx | DDMMMYYYY/Hh:mm | XXXXX/XXXXX | | | | |
| | CONTRACTOR OF | XXXX | DDMMMYYYY/Hh:mm | | | | | |
| | | XXXX | DDMMMYYYY/Hh:mm | | | | | |
| | | XXXX | DDMMMYYYY/Hh:mm | | | | | |
| | | Day -1 | | | | | | |
| | | Mean Use | | | | | | |

| Footnotes: | For the purpose of this listing one month is assumed to have 30 days. |
|---|---|
| | Duration of period and event rate will only be calculated if the visit at the end of the reporting period took place. |
| Programming Notes : | [1] As required to be modified based on data and any applicable IDSL standard principles for listings |
| | [2] If all units are IU or convertible to IU combine Dose and Unit columns to a single Column Dose (IU) |

OTX116505

Example: OTHER\_L7 Protocol : OTX116505

Protocol: OTX116505
Population: Safety


### Listing XX Cardiovascular Events

| XXXXX Male/White Pulmonary Hypertens. | | Inv./ | Age(yrs)/<br>Sex/ | 771 - 1 - | Data | Cardiovascular | Proceeding. |
|---|---|---|---|---|---|---|---|
| XXXXX/ 27/ XXX DDMMMYYYY Yes Congestive Heart Fai. XXXXX Male/ White Pulmonary Hypertens. | reatment | Subj. | Race | VISIT | Date | | Events |
| XXXXX XXXXX/ 27/ XXX DDMMMYYYY Yes Congestive Heart Fai. XXXXX Male/ White Pulmonary Hypertens. | | | | | | No | |
| Pulmonary Hypertens | xxxx | | Male/ | XXX | DDMMMYYYY | Yes | Congestive Heart Failure |
| | | | | | | | Pulmonary Hypertension |
| No | | | | | | No | |


Protocol : OTX116505 Population : Safety

# Listing XX Listing of C-Peptide & Glucose from Clamp

Treatment:Placebo

| | | | | | Planned/Actua | al | Glucose<br>Infusion | | |
|---|---|---|---|---|---|---|---|---|---|
| | Age(yrs)/ | | | | Relative | Time | Concentration | | |
| Inv./ | Sex/ | | Date/ | | Time | Sample | and Rate | C-Peptide | Glucose |
| Subj. | Race | Visit | Study Day | Phase | (Mins) | Taken | (ml/hr). | (Units) | (Units) |
| XXXXX/<br>XXX | XX/<br>Male/<br>White | XXXX | DDMMMYYYY / XX | Euglycemic | X/X | HH:MM | Gluc 10%,<br>50ml/hr | XXX.XX | XXX.XX |
| | vviiite | | | | Χ | HH:MM | Gluc 20%, 100<br>ml/hr | XXX.XX | XXX.XX |
| | | | | Hyperglycemic | X | HH:MM | NaCl, 50 ml/hr | XXX.XX | XXX.XX |
| | | | | 21 07 | X | HH:MM | | XXX.XX | XXX.XX |
| | | | | | X | HH:MM | | XXX.XX | XXX.XX |
| | | XXXX | DDMMMYYYY/XX | | Х | HH:MM | | XXX.XX | XXX.XX |
| | | | | | X | HH:MM | | XXX.XX | XXX.XX |
| | | | | | X | HH:MM | | XXX.XX | XXX.XX |

| The second secon | |
|---|---|
| Programming Notes : | [1] As required to be modified based on data and any applicable IDSL standard principles for listings |

OTX116505


Protocol: OTX116505 Population : Safety

Listing XX
Listing of C-Peptide & Glucose from Clamp: Derived Parameters

#### Treatment: Placebo

| Inv./ | | | | Time Int. For<br>Derivation | | Change |
|---|---|---|---|---|---|---|
| Subj. | Parameter | Visit | Date/Study Day | (Mins) | Result | from Baseline |
| XXXXX/<br>XXX | Glucose Weighted<br>Mean AUC(60-140M)<br>(UNIT) | XXXX | DDMMMYYYY / XX | XXX | X.XXX | X.XXX |
| | (ONT) | XXXX | | XXX | X.XXX | X.XXX |
| | | XXXX | | XXX | X.XXX | X.XXX |
| | | XXXX | | XXX | X.XXX | X.XXX |
| | XXXX | XXXX | | | X.XXX | X.XXX |
| | | XXXX | | | X.XXX | X.XXX |
| | | XXXX | | | X.XXX | X.XXX |
| | | XXXX | | | X.XXX | X.XXX |

| Programming Notes : | [1] As required to be modified based on data and any applicable IDSL standard principles for listings |
|---|---|
| (20) | [2] Include the following parameters: Glucose weighted mean (60-140), C-Peptide weighted mean (60-140), Insulin Sensitivity |

Example : OTHER\_L10

Protocol : OTX116505 Population : Safety Page 1 of X

Listing XX

Listing of Family History of Cardiovascular Risk

Treatment: Placebo

| Inv./<br>Subj. | Family History<br>Classification | Family History<br>Relative | Family History of<br>Premature Coronary<br>Disease |
|---|---|---|---|
| XXXXX/ | Cardiovascular Risk | First Degree | |
| XXX | Factor | Relative | |

Footnote

Premature is defined when occurring before 65 years in women or before 55 years in men. Only first degree relatives are considered.

OTX116505

Example : OTHER\_L11

Protocol : OTX116505
Population : Safety

Listing XX
Listing of Substance Use


Treatment: Placebo

| Inv./ | History of Smoking | Date of Last | Alcohol | Average Number of |
|---|---|---|---|---|
| Subj. | Status | Smoking | Consumption | Units |
| XXXXX/<br>XXX | Former smoker | DDMMMYYYY | | |

Footnote Premature is defined when occurring before 65 years in women or before 55 years in men. Only first degree relatives are considered.


Protocol : OTX116505 Population : Safety

**Listing XX** 

| | Age(yrs)/<br>Sex/ | | | | | Change from |
|---|---|---|---|---|---|---|
| Inv./Subj. | Race | Visit | Date/Study Day | Test (Unit) | Result | Baseline |
| XXXXX/ XXX | XX/ | XXXX | | | | |
| | Male/ | | DDMMMYYYY / XX | | | |
| | White | | | | | |
| | | XXXX | | | | |
| | | XXXX | | | | |
| | | XXXX | | | | |
| | | XXXX | | | | |
| | | XXXX | | | | |
| | | XXXX | | | | |
| | | XXXX | | | | |

Programming Notes: [1] As required to be modified based on data and any applicable IDSL standard principles for listings

### **PAREXEL International Electronic Signature Page**

This page is the manifestation of the electronic signature(s) used in compliance with PAREXEL International's electronic signature policies and procedures and in compliance with applicable regulations.

UserName: PPD

Title: Senior Biostatistician, GDO

Date: Tuesday, 20 November 2018, 02:26 PM GMT Standard Time

Meaning: Document contents approved.

\_\_\_\_\_